CLINICAL TRIAL: NCT01289990
Title: A Phase III Double-blind, Extension, Placebo-controlled Parallel Group Safety and Efficacy Trial of BI 10773 (10 and 25mg Once Daily) and Sitagliptin (100mg Once Daily) Given for Minimum 76 Weeks (Incl. 24 Weeks of Preceding Trial) as Monotherapy or With Different Back-ground Therapies in Patients With Type 2 Diabetes Mellitus Previously Completing Trial 1245.19, 1245.20 or 1245.23
Brief Title: Safety and Efficacy of Empagliflozin (BI 10773) and Sitagliptin Versus Placebo Over 76 Weeks in Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1245.31; 2010-022718-17 (EudraCT Number: EudraCT)
Record Dates: First submitted 2011-01-31; First posted 2011-02-04 (Estimated); Results first posted 2014-07-15 (Estimated); Last update posted 2014-07-15 (Estimated); Status verified 2014-07

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — empagliflozin; Sitagliptin Phosphate

ARMS (13):
- BI 10773 low (drug naive) (Experimental): BI 10773 tablets once daily
  Interventions: Drug: BI 10773; Drug: Placebo
- BI 10773 high (drug naive) (Experimental): BI 10773 tablets once daily
  Interventions: Drug: Placebo; Drug: BI 10773
- Placebo (drug naive) (Placebo Comparator): Placebo tablets matching BI 10773 / Sitagliptin once daily
  Interventions: Drug: Placebo
- Sitagliptin 100mg (drug naive) (Active Comparator): Sitagliptin once daily
  Interventions: Drug: Placebo; Drug: Sitagliptin 100mg
- BI 10773 low (pioglitazone) (Experimental): BI 10773 tablets once daily
  Interventions: Drug: BI 10773; Drug: Placebo
- BI 10773 high (pioglitazone) (Experimental): BI 10773 tablets once daily
  Interventions: Drug: BI 10773; Drug: Placebo
- Placebo (pioglitazone) (Placebo Comparator): Placebo tablets matching BI 10773 once daily
  Interventions: Drug: Placebo
- BI 10773 low (metformin) (Experimental): BI 10773 tablets once daily
  Interventions: Drug: Placebo; Drug: BI 10773
- BI 10773 high (metformin) (Experimental): BI 10773 tablets once daily
  Interventions: Drug: BI 10773; Drug: Placebo
- Placebo (metformin) (Placebo Comparator): Placebo tablets matching BI 10773 once daily
  Interventions: Drug: Placebo
- BI 10773 low (metformin+sulfonylurea) (Experimental): BI 10773 tablets once daily
  Interventions: Drug: BI 10773; Drug: Placebo
- BI 10773 high (metformin+sulfonylurea) (Experimental): BI 10773 tablets once daily
  Interventions: Drug: BI 10773; Drug: Placebo
- Placebo (metformin+sulfonylurea) (Placebo Comparator): Placebo tablets matching BI 10773
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BI 10773 — BI 10773 tablets once daily
  Arms: BI 10773 low (drug naive)
Drug: Placebo — Placebo matching BI 10773 low dose
  Arms: Placebo (drug naive)
Drug: Placebo — Placebo matching BI 10773 high dose
  Arms: Sitagliptin 100mg (drug naive)
Drug: Placebo — Placebo matching Sitagliptin
  Arms: Placebo (drug naive)
Drug: Placebo — Placebo matching BI 10773 high dose
  Arms: BI 10773 low (metformin)
Drug: Placebo — Placebo matching BI 10773 high dose
  Arms: Placebo (drug naive)
Drug: BI 10773 — BI 10773 tablets once daily
  Arms: BI 10773 high (metformin)
Drug: Placebo — Placebo matching BI 10773 low dose
  Arms: Placebo (pioglitazone)
Drug: Placebo — Placebo matching BI 10773 low dose
  Arms: Sitagliptin 100mg (drug naive)
Drug: BI 10773 — BI 10773 tablets once daily
  Arms: BI 10773 low (pioglitazone)
Drug: Placebo — Placebo matching BI 10773 low dose
  Arms: Placebo (metformin)
Drug: Placebo — Placebo matching BI 10773 high dose
  Arms: BI 10773 low (pioglitazone)
Drug: Placebo — Placebo matching Sitagliptin
  Arms: BI 10773 high (drug naive)
Drug: BI 10773 — BI 10773 tablets once daily
  Arms: BI 10773 low (metformin)
Drug: BI 10773 — BI 10773 tablets once daily
  Arms: BI 10773 low (metformin+sulfonylurea)
Drug: BI 10773 — BI 10773 tablets once daily
  Arms: BI 10773 high (drug naive)
Drug: Placebo — Placebo matching BI 10773 high dose
  Arms: Placebo (metformin)
Drug: BI 10773 — BI 10773 tablets once daily
  Arms: BI 10773 high (metformin+sulfonylurea)
Drug: Placebo — Placebo matching BI 10773 low dose
  Arms: BI 10773 high (metformin+sulfonylurea)
Drug: Placebo — Placebo matching BI 10773 high dose
  Arms: Placebo (pioglitazone)
Drug: Placebo — Placebo matching Sitagliptin
  Arms: BI 10773 low (drug naive)
Drug: Sitagliptin 100mg — Sitagliptin once daily
  Arms: Sitagliptin 100mg (drug naive)
Drug: BI 10773 — BI 10773 tablets once daily
  Arms: BI 10773 high (pioglitazone)
Drug: Placebo — Placebo matching BI 10773 low dose
  Arms: BI 10773 high (pioglitazone)
Drug: Placebo — Placebo matching BI 10773 low dose
  Arms: Placebo (metformin+sulfonylurea)
Drug: Placebo — Placebo matching BI 10773 low dose
  Arms: BI 10773 high (drug naive)
Drug: Placebo — Placebo matching BI 10773 high dose
  Arms: Placebo (metformin+sulfonylurea)
Drug: Placebo — Placebo matching BI 10773 low dose
  Arms: BI 10773 high (metformin)
Drug: Placebo — Placebo matching BI 10773 high dose
  Arms: BI 10773 low (metformin+sulfonylurea)
Drug: Placebo — Placebo matching BI 10773 high dose
  Arms: BI 10773 low (drug naive)

SUMMARY:
This study will investigate the efficacy and long term safety and tolerability of BI 10773 in type 2 diabetic patients.

ELIGIBILITY:
Inclusion criteria:

1. Patients completing the entire treatment period of the preceding double-blind trial 1245.19, 1245.20 or 1245.23 with or without rescue therapy.
2. Signed and dated written informed consent by date of Visit 1 in accordance with Good Clinical Practice and local legislation.

Exclusion criteria:

1. Patient who meet one or more of the withdrawal criteria of the treatment period of the previous trial 1245.19, 1245.20 or 1245.23.
2. Indication of liver disease, defined by serum levels of either alanine aminotransferase , aspartate aminotransferase, or alkaline phosphatase above 3 x upper limit of normal as determined during last visit of preceding trial.
3. Impaired renal function defined as glomerular filtration rate<30 ml/min (severe renal impairment, Modification of Diet in Renal Disease formula) as determined during last visit of preceding trial.
4. Contraindications to sitagliptin, pioglitazone, metformin or sulfonylurea according to local label, which started during trial participation in 1245.19, 1245.20 or 1245.23
5. Pre-menopausal women (last menstruation < or = 1 year prior to informed consent) who are nursing or pregnant or are of child-bearing potential and are not practicing an acceptable method of birth control, or do not plan to continue using this method throughout the study and do not agree to submit to periodic pregnancy testing during participation in the trial. Acceptable methods of birth control include tubal ligation, transdermal patch, intra uterine devices/systems, oral, implantable or injectable contraceptives, sexual abstinence (if acceptable by local authorities), double barrier method and vasectomised partner.
6. Alcohol or drug abuse within the 3 months prior to informed consent that would interfere with trial participation or any ongoing condition leading to a decreased compliance to study procedures or study drug intake.
7. Participation in another trial with an investigational drug within 30 days prior to informed consent (except 1245.19, 1245.20 and 1245.23).
8. Any other clinical condition that would jeopardize patient's safety while participating in this clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2705 (Actual)
Dates: Start 2011-02; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (243):
- United States (40):
  - 1245.31.10145 Boehringer Ingelheim Investigational Site, Birmingham, Alabama
  - 1245.31.10162 Boehringer Ingelheim Investigational Site, Glendale, Arizona
  - 1245.31.10124 Boehringer Ingelheim Investigational Site, Mesa, Arizona
  - 1245.31.10108 Boehringer Ingelheim Investigational Site, Phoenix, Arizona
  - 1245.31.10046 Boehringer Ingelheim Investigational Site, Tempe, Arizona
  - 1245.31.10154 Boehringer Ingelheim Investigational Site, Chino, California
  - 1245.31.10149 Boehringer Ingelheim Investigational Site, Rancho Cucamonga, California
  - 1245.31.10131 Boehringer Ingelheim Investigational Site, West Hills, California
  - 1245.31.10038 Boehringer Ingelheim Investigational Site, Northglenn, Colorado
  - 1245.31.10127 Boehringer Ingelheim Investigational Site, Waterbury, Connecticut
  - 1245.31.10137 Boehringer Ingelheim Investigational Site, Clearwater, Florida
  - 1245.31.10133 Boehringer Ingelheim Investigational Site, Jupiter, Florida
  - 1245.31.10006 Boehringer Ingelheim Investigational Site, Miami, Florida
  - 1245.31.10085 Boehringer Ingelheim Investigational Site, Plantation, Florida
  - 1245.31.10080 Boehringer Ingelheim Investigational Site, Decatur, Georgia
  - 1245.31.10077 Boehringer Ingelheim Investigational Site, Perry, Georgia
  - 1245.31.10001 Boehringer Ingelheim Investigational Site, Chicago, Illinois
  - 1245.31.10159 Boehringer Ingelheim Investigational Site, Des Moines, Iowa
  - 1245.31.10014 Boehringer Ingelheim Investigational Site, Dubuque, Iowa
  - 1245.31.10117 Boehringer Ingelheim Investigational Site, Arkansas City, Kansas
  - 1245.31.10157 Boehringer Ingelheim Investigational Site, Newton, Kansas
  - 1245.31.10146 Boehringer Ingelheim Investigational Site, Louisville, Kentucky
  - 1245.31.10003 Boehringer Ingelheim Investigational Site, Dearborn, Michigan
  - 1245.31.10059 Boehringer Ingelheim Investigational Site, New Hyde Park, New York
  - 1245.31.10034 Boehringer Ingelheim Investigational Site, Rochester, New York
  - 1245.31.10123 Boehringer Ingelheim Investigational Site, Smithtown, New York
  - 1245.31.10071 Boehringer Ingelheim Investigational Site, Asheboro, North Carolina
  - 1245.31.10086 Boehringer Ingelheim Investigational Site, Salisbury, North Carolina
  - 1245.31.10129 Boehringer Ingelheim Investigational Site, Carlisle, Ohio
  - 1245.31.10045 Boehringer Ingelheim Investigational Site, Cincinnati, Ohio
  - 1245.31.10119 Boehringer Ingelheim Investigational Site, Cincinnati, Ohio
  - 1245.31.10130 Boehringer Ingelheim Investigational Site, Gallipolis, Ohio
  - 1245.31.10158 Boehringer Ingelheim Investigational Site, Mt. Pleasant, South Carolina
  - 1245.31.10015 Boehringer Ingelheim Investigational Site, Simpsonville, South Carolina
  - 1245.31.10033 Boehringer Ingelheim Investigational Site, Chattanooga, Tennessee
  - 1245.31.10112 Boehringer Ingelheim Investigational Site, Memphis, Tennessee
  - 1245.31.10156 Boehringer Ingelheim Investigational Site, Houston, Texas
  - 1245.31.10151 Boehringer Ingelheim Investigational Site, Hurst, Texas
  - 1245.31.10143 Boehringer Ingelheim Investigational Site, Killeen, Texas
  - 1245.31.10155 Boehringer Ingelheim Investigational Site, San Antonio, Texas
- Belgium (12):
  - 1245.31.32008 Boehringer Ingelheim Investigational Site, Brussels
  - 1245.31.32023 Boehringer Ingelheim Investigational Site, Brussels
  - 1245.31.32003 Boehringer Ingelheim Investigational Site, De Pinte
  - 1245.31.32015 Boehringer Ingelheim Investigational Site, Deurne
  - 1245.31.32016 Boehringer Ingelheim Investigational Site, Deurne
  - 1245.31.32025 Boehringer Ingelheim Investigational Site, Gozée
  - 1245.31.32019 Boehringer Ingelheim Investigational Site, Leopoldsburg
  - 1245.31.32024 Boehringer Ingelheim Investigational Site, Linkebeek
  - 1245.31.32021 Boehringer Ingelheim Investigational Site, Mouscron
  - 1245.31.32020 Boehringer Ingelheim Investigational Site, Sint-Gillis-Waas
  - 1245.31.32018 Boehringer Ingelheim Investigational Site, Tielt
  - 1245.31.32026 Boehringer Ingelheim Investigational Site, Tremelo
- Canada (35):
  - 1245.31.20032 Boehringer Ingelheim Investigational Site, Calgary, Alberta
  - 1245.31.20023 Boehringer Ingelheim Investigational Site, Edmonton, Alberta
  - 1245.31.20011 Boehringer Ingelheim Investigational Site, Chilliwack, British Columbia
  - 1245.31.20028 Boehringer Ingelheim Investigational Site, Vancouver, British Columbia
  - 1245.31.20018 Boehringer Ingelheim Investigational Site, Victoria, British Columbia
  - 1245.31.20033 Boehringer Ingelheim Investigational Site, Victoria, British Columbia
  - 1245.31.20015 Boehringer Ingelheim Investigational Site, Winnipeg, Manitoba
  - 1245.31.20012 Boehringer Ingelheim Investigational Site, Moncton, New Brunswick
  - 1245.31.20016 Boehringer Ingelheim Investigational Site, Mount Pearl, Newfoundland and Labrador
  - 1245.31.20024 Boehringer Ingelheim Investigational Site, Paradise, Newfoundland and Labrador
  - 1245.31.20008 Boehringer Ingelheim Investigational Site, St. John's, Newfoundland and Labrador
  - 1245.31.20026 Boehringer Ingelheim Investigational Site, Halifax, Nova Scotia
  - 1245.31.20022 Boehringer Ingelheim Investigational Site, Brampton, Ontario
  - 1245.31.20057 Boehringer Ingelheim Investigational Site, Brampton, Ontario
  - 1245.31.20035 Boehringer Ingelheim Investigational Site, Corunna, Ontario
  - 1245.31.20030 Boehringer Ingelheim Investigational Site, Etobicoke, Ontario
  - 1245.31.20019 Boehringer Ingelheim Investigational Site, Hamilton, Ontario
  - 1245.31.20017 Boehringer Ingelheim Investigational Site, London, Ontario
  - 1245.31.20029 Boehringer Ingelheim Investigational Site, London, Ontario
  - 1245.31.20060 Boehringer Ingelheim Investigational Site, London, Ontario
  - 1245.31.20003 Boehringer Ingelheim Investigational Site, Markham, Ontario
  - 1245.31.20009 Boehringer Ingelheim Investigational Site, Newmarket, Ontario
  - 1245.31.20040 Boehringer Ingelheim Investigational Site, Oakville, Ontario
  - 1245.31.20034 Boehringer Ingelheim Investigational Site, Sarnia, Ontario
  - 1245.31.20005 Boehringer Ingelheim Investigational Site, Strathroy, Ontario
  - 1245.31.20002 Boehringer Ingelheim Investigational Site, Toronto, Ontario
  - 1245.31.20006 Boehringer Ingelheim Investigational Site, Toronto, Ontario
  - 1245.31.20007 Boehringer Ingelheim Investigational Site, Montague, Prince Edward Island
  - 1245.31.20027 Boehringer Ingelheim Investigational Site, Laval, Quebec
  - 1245.31.20025 Boehringer Ingelheim Investigational Site, Montreal, Quebec
  - 1245.31.20058 Boehringer Ingelheim Investigational Site, Saint Romuald, Quebec
  - 1245.31.20038 Boehringer Ingelheim Investigational Site, Saint-Laurent, Quebec
  - 1245.31.20036 Boehringer Ingelheim Investigational Site, Sherbrooke, Quebec
  - 1245.31.20021 Boehringer Ingelheim Investigational Site, Trois-Rivières, Quebec
  - 1245.31.20041 Boehringer Ingelheim Investigational Site, Saskatoon, Saskatchewan
- China (35):
  - 1245.31.86007 Boehringer Ingelheim Investigational Site, Beijing
  - 1245.31.86008 Boehringer Ingelheim Investigational Site, Beijing
  - 1245.31.86031 Boehringer Ingelheim Investigational Site, Beijing
  - 1245.31.86032 Boehringer Ingelheim Investigational Site, Beijing
  - 1245.31.86033 Boehringer Ingelheim Investigational Site, Beijing
  - 1245.31.86034 Boehringer Ingelheim Investigational Site, Beijing
  - 1245.31.86035 Boehringer Ingelheim Investigational Site, Beijing
  - 1245.31.86058 Boehringer Ingelheim Investigational Site, Chongqing
  - 1245.31.86038 Boehringer Ingelheim Investigational Site, Dalian
  - 1245.31.86001 Boehringer Ingelheim Investigational Site, Guangzhou
  - 1245.31.86003 Boehringer Ingelheim Investigational Site, Guangzhou
  - 1245.31.86052 Boehringer Ingelheim Investigational Site, Guangzhou
  - 1245.31.86012 Boehringer Ingelheim Investigational Site, Guiyang
  - 1245.31.86037 Boehringer Ingelheim Investigational Site, Haerbin
  - 1245.31.86020 Boehringer Ingelheim Investigational Site, Hangzhou
  - 1245.31.86049 Boehringer Ingelheim Investigational Site, Jinan
  - 1245.31.86053 Boehringer Ingelheim Investigational Site, Jinan
  - 1245.31.86018 Boehringer Ingelheim Investigational Site, Jingzhou
  - 1245.31.86019 Boehringer Ingelheim Investigational Site, Nanchang
  - 1245.31.86042 Boehringer Ingelheim Investigational Site, Nanjing
  - 1245.31.86043 Boehringer Ingelheim Investigational Site, Nanjing
  - 1245.31.86055 Boehringer Ingelheim Investigational Site, Nanning
  - 1245.31.86056 Boehringer Ingelheim Investigational Site, Nanning
  - 1245.31.86016 Boehringer Ingelheim Investigational Site, Qingdao
  - 1245.31.86039 Boehringer Ingelheim Investigational Site, Shanghai
  - 1245.31.86054 Boehringer Ingelheim Investigational Site, Shantou
  - 1245.31.86057 Boehringer Ingelheim Investigational Site, Shenyang
  - 1245.31.86045 Boehringer Ingelheim Investigational Site, Shijiazhuang
  - 1245.31.86017 Boehringer Ingelheim Investigational Site, Shiyan
  - 1245.31.86013 Boehringer Ingelheim Investigational Site, Suzhou
  - 1245.31.86015 Boehringer Ingelheim Investigational Site, Taiyuan
  - 1245.31.86036 Boehringer Ingelheim Investigational Site, Tianjin
  - 1245.31.86011 Boehringer Ingelheim Investigational Site, Xi'an
  - 1245.31.86041 Boehringer Ingelheim Investigational Site, Xi'an
  - 1245.31.86014 Boehringer Ingelheim Investigational Site, Xiamen
- France (15):
  - 1245.31.33008 Boehringer Ingelheim Investigational Site, Bersée
  - 1245.31.33020 Boehringer Ingelheim Investigational Site, Bischheim
  - 1245.31.33002 Boehringer Ingelheim Investigational Site, Bondy
  - 1245.31.33016 Boehringer Ingelheim Investigational Site, Bruay-la-Buissière
  - 1245.31.33001 Boehringer Ingelheim Investigational Site, Corbeil-Essonnes
  - 1245.31.33010 Boehringer Ingelheim Investigational Site, Croix
  - 1245.31.33009 Boehringer Ingelheim Investigational Site, Hautmont
  - 1245.31.33003 Boehringer Ingelheim Investigational Site, La Rochelle
  - 1245.31.33045 Boehringer Ingelheim Investigational Site, Marseille
  - 1245.31.33004 Boehringer Ingelheim Investigational Site, Narbonne
  - 1245.31.33012 Boehringer Ingelheim Investigational Site, Schiltigheim
  - 1245.31.33013 Boehringer Ingelheim Investigational Site, Strasbourg
  - 1245.31.33019 Boehringer Ingelheim Investigational Site, Strasbourg
  - 1245.31.33007 Boehringer Ingelheim Investigational Site, Vieux-Condé
  - 1245.31.33018 Boehringer Ingelheim Investigational Site, Wattrelos
- Germany (18):
  - 1245.31.49001 Boehringer Ingelheim Investigational Site, Dormagen
  - 1245.31.49013 Boehringer Ingelheim Investigational Site, Dresden
  - 1245.31.49016 Boehringer Ingelheim Investigational Site, Düsseldorf
  - 1245.31.49009 Boehringer Ingelheim Investigational Site, Flörsheim
  - 1245.31.49015 Boehringer Ingelheim Investigational Site, Frankfurt
  - 1245.31.49019 Boehringer Ingelheim Investigational Site, Haag
  - 1245.31.49004 Boehringer Ingelheim Investigational Site, Hatten
  - 1245.31.49020 Boehringer Ingelheim Investigational Site, Hohenmölsen
  - 1245.31.49007 Boehringer Ingelheim Investigational Site, Künzing
  - 1245.31.49002 Boehringer Ingelheim Investigational Site, Neuwied
  - 1245.31.49008 Boehringer Ingelheim Investigational Site, Nuremberg
  - 1245.31.49010 Boehringer Ingelheim Investigational Site, Rednitzhembach
  - 1245.31.49006 Boehringer Ingelheim Investigational Site, Rehburg-Loccum
  - 1245.31.49011 Boehringer Ingelheim Investigational Site, Rehlingen-Siersburg
  - 1245.31.49005 Boehringer Ingelheim Investigational Site, Saarbrücken
  - 1245.31.49017 Boehringer Ingelheim Investigational Site, Saint Ingbert/Oberwürzbach
  - 1245.31.49022 Boehringer Ingelheim Investigational Site, Schauenburg
  - 1245.31.49003 Boehringer Ingelheim Investigational Site, Unterschneidheim
- 1245.31.30004 Boehringer Ingelheim Investigational Site, Thessaloniki, Greece
- India (17):
  - 1245.31.91005 Boehringer Ingelheim Investigational Site, Bangalore
  - 1245.31.91006 Boehringer Ingelheim Investigational Site, Bangalore
  - 1245.31.91008 Boehringer Ingelheim Investigational Site, Bangalore
  - 1245.31.91003 Boehringer Ingelheim Investigational Site, Belagavi
  - 1245.31.91004 Boehringer Ingelheim Investigational Site, Chennai
  - 1245.31.91009 Boehringer Ingelheim Investigational Site, Chennai
  - 1245.31.91001 Boehringer Ingelheim Investigational Site, Coimbatore
  - 1245.31.91101 Boehringer Ingelheim Investigational Site, Coimbatore
  - 1245.31.91104 Boehringer Ingelheim Investigational Site, Indore
  - 1245.31.91015 Boehringer Ingelheim Investigational Site, Kalaburagi
  - 1245.31.91103 Boehringer Ingelheim Investigational Site, Maharashtra
  - 1245.31.91002 Boehringer Ingelheim Investigational Site, Mumbai
  - 1245.31.91007 Boehringer Ingelheim Investigational Site, Mumbai, Maharastra
  - 1245.31.91010 Boehringer Ingelheim Investigational Site, Nagpur
  - 1245.31.91012 Boehringer Ingelheim Investigational Site, New Delhi
  - 1245.31.91014 Boehringer Ingelheim Investigational Site, Pune
  - 1245.31.91105 Boehringer Ingelheim Investigational Site, Pune
- Ireland (5):
  - 1245.31.35304 Boehringer Ingelheim Investigational Site, Birr, Co. Offaly
  - 1245.31.35302 Boehringer Ingelheim Investigational Site, Co. Cork
  - 1245.31.35305 Boehringer Ingelheim Investigational Site, Co. Galway
  - 1245.31.35303 Boehringer Ingelheim Investigational Site, Co. Wexford
  - 1245.31.35306 Boehringer Ingelheim Investigational Site, Co. Wexford
- Japan (12):
  - 1245.31.81007 Boehringer Ingelheim Investigational Site, Chiyoda-ku, Tokyo
  - 1245.31.81001 Boehringer Ingelheim Investigational Site, Chuo-ku, Tokyo
  - 1245.31.81002 Boehringer Ingelheim Investigational Site, Chuo-ku, Tokyo
  - 1245.31.81005 Boehringer Ingelheim Investigational Site, Ebetsu, Hokkaido
  - 1245.31.81004 Boehringer Ingelheim Investigational Site, Kamakura, Kanagawa
  - 1245.31.81003 Boehringer Ingelheim Investigational Site, Minato-ku, Tokyo
  - 1245.31.81006 Boehringer Ingelheim Investigational Site, Shinjuku-ku, Tokyo
  - 1245.31.81008 Boehringer Ingelheim Investigational Site, Shinjuku-ku, Tokyo
  - 1245.31.81009 Boehringer Ingelheim Investigational Site, Suita, Osaka
  - 1245.31.81010 Boehringer Ingelheim Investigational Site, Ube, Yamaguchi
  - 1245.31.81012 Boehringer Ingelheim Investigational Site, Urasoe, Okinawa
  - 1245.31.81013 Boehringer Ingelheim Investigational Site, Urasoe, Okinawa
- Mexico (4):
  - 1245.31.52003 Boehringer Ingelheim Investigational Site, Guadalajara
  - 1245.31.52004 Boehringer Ingelheim Investigational Site, Guadalajara
  - 1245.31.52001 Boehringer Ingelheim Investigational Site, Monterrey
  - 1245.31.52002 Boehringer Ingelheim Investigational Site, Monterrey
- Philippines (5):
  - 1245.31.63002 Boehringer Ingelheim Investigational Site, Cebu
  - 1245.31.63003 Boehringer Ingelheim Investigational Site, Davao City
  - 1245.31.63001 Boehringer Ingelheim Investigational Site, Manila
  - 1245.31.63004 Boehringer Ingelheim Investigational Site, Manila
  - 1245.31.63005 Boehringer Ingelheim Investigational Site, Manila
- Slovakia (7):
  - 1245.31.74005 Boehringer Ingelheim Investigational Site, Bratislava
  - 1245.31.74002 Boehringer Ingelheim Investigational Site, Lučenec
  - 1245.31.74006 Boehringer Ingelheim Investigational Site, Nitra
  - 1245.31.74014 Boehringer Ingelheim Investigational Site, Nové Zámky
  - 1245.31.74001 Boehringer Ingelheim Investigational Site, Považská Bystrica
  - 1245.31.74004 Boehringer Ingelheim Investigational Site, Prešov
  - 1245.31.74003 Boehringer Ingelheim Investigational Site, Trebišov
- Slovenia (3):
  - 1245.31.38003 Boehringer Ingelheim Investigational Site, Celje
  - 1245.31.38002 Boehringer Ingelheim Investigational Site, Koper
  - 1245.31.38001 Boehringer Ingelheim Investigational Site, Maribor
- South Korea (13):
  - 1245.31.82012 Boehringer Ingelheim Investigational Site, Anyang
  - 1245.31.82011 Boehringer Ingelheim Investigational Site, Goyang
  - 1245.31.82009 Boehringer Ingelheim Investigational Site, Ilsan
  - 1245.31.82001 Boehringer Ingelheim Investigational Site, Incheon
  - 1245.31.82006 Boehringer Ingelheim Investigational Site, Jeonju
  - 1245.31.82004 Boehringer Ingelheim Investigational Site, Pusan
  - 1245.31.82005 Boehringer Ingelheim Investigational Site, Seoul
  - 1245.31.82007 Boehringer Ingelheim Investigational Site, Seoul
  - 1245.31.82008 Boehringer Ingelheim Investigational Site, Seoul
  - 1245.31.82010 Boehringer Ingelheim Investigational Site, Seoul
  - 1245.31.82014 Boehringer Ingelheim Investigational Site, Seoul
  - 1245.31.82002 Boehringer Ingelheim Investigational Site, Suwon
  - 1245.31.82003 Boehringer Ingelheim Investigational Site, Wŏnju
- Switzerland (2):
  - 1245.31.41004 Boehringer Ingelheim Investigational Site, Lugano
  - 1245.31.41003 Boehringer Ingelheim Investigational Site, Rorschach
- Taiwan (9):
  - 1245.31.88010 Boehringer Ingelheim Investigational Site, Kaohsiung City
  - 1245.31.88011 Boehringer Ingelheim Investigational Site, Kaohsiung City
  - 1245.31.88012 Boehringer Ingelheim Investigational Site, Kaohsiung City
  - 1245.31.88013 Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - 1245.31.88009 Boehringer Ingelheim Investigational Site, Taichung
  - 1245.31.88014 Boehringer Ingelheim Investigational Site, Tainan
  - 1245.31.88006 Boehringer Ingelheim Investigational Site, Taipei
  - 1245.31.88021 Boehringer Ingelheim Investigational Site, Taipei
  - 1245.31.88008 Boehringer Ingelheim Investigational Site, Taoyuan
- Turkey (Türkiye) (5):
  - 1245.31.90003 Boehringer Ingelheim Investigational Site, Erzurum
  - 1245.31.90001 Boehringer Ingelheim Investigational Site, Gaziantep
  - 1245.31.90002 Boehringer Ingelheim Investigational Site, Istanbul
  - 1245.31.90006 Boehringer Ingelheim Investigational Site, Istanbul
  - 1245.31.90004 Boehringer Ingelheim Investigational Site, Izmir
- Ukraine (5):
  - 1245.31.75002 Boehringer Ingelheim Investigational Site, Dnipro
  - 1245.31.75001 Boehringer Ingelheim Investigational Site, Kharkiv
  - 1245.31.75006 Boehringer Ingelheim Investigational Site, Lviv
  - 1245.31.75004 Boehringer Ingelheim Investigational Site, Vinnitsa
  - 1245.31.75003 Boehringer Ingelheim Investigational Site, Vinnytsia

REFERENCES:
- [Derived] Tuttle KR, Levin A, Nangaku M, Kadowaki T, Agarwal R, Hauske SJ, Elsasser A, Ritter I, Steubl D, Wanner C, Wheeler DC. Safety of Empagliflozin in Patients With Type 2 Diabetes and Chronic Kidney Disease: Pooled Analysis of Placebo-Controlled Clinical Trials. Diabetes Care. 2022 Jun 2;45(6):1445-1452. doi: 10.2337/dc21-2034. PMID 35472672
- [Derived] Inzucchi SE, Davies MJ, Khunti K, Trivedi P, George JT, Zwiener I, Johansen OE, Sattar N. Empagliflozin treatment effects across categories of baseline HbA1c, body weight and blood pressure as an add-on to metformin in patients with type 2 diabetes. Diabetes Obes Metab. 2021 Feb;23(2):425-433. doi: 10.1111/dom.14234. Epub 2020 Nov 20. PMID 33084149
- [Derived] Shiba T, Ishii S, Okamura T, Mitsuyoshi R, Pfarr E, Koiwai K. Efficacy and safety of empagliflozin in Japanese patients with type 2 diabetes mellitus: A sub-analysis by body mass index and age of pooled data from three clinical trials. Diabetes Res Clin Pract. 2017 Sep;131:169-178. doi: 10.1016/j.diabres.2017.07.004. Epub 2017 Jul 8. PMID 28753486
- [Derived] Roden M, Merker L, Christiansen AV, Roux F, Salsali A, Kim G, Stella P, Woerle HJ, Broedl UC; EMPA-REG EXTEND MONO investigators. Safety, tolerability and effects on cardiometabolic risk factors of empagliflozin monotherapy in drug-naive patients with type 2 diabetes: a double-blind extension of a Phase III randomized controlled trial. Cardiovasc Diabetol. 2015 Dec 23;14:154. doi: 10.1186/s12933-015-0314-0. PMID 26701110
- [Derived] Haering HU, Merker L, Christiansen AV, Roux F, Salsali A, Kim G, Meinicke T, Woerle HJ, Broedl UC; EMPA-REG EXTEND METSU investigators. Empagliflozin as add-on to metformin plus sulphonylurea in patients with type 2 diabetes. Diabetes Res Clin Pract. 2015 Oct;110(1):82-90. doi: 10.1016/j.diabres.2015.05.044. Epub 2015 May 29. PMID 26324220

RESULTS

PARTICIPANT FLOW:
Groups:
- Empagliflozin 10 mg (Drug Naive): Patients rolled over from trial 1245.20
  Empagliflozin 10 mg tablets once daily
  Placebo: Placebo matching Sitagliptin
  Placebo: Placebo matching Empagliflozin 25 mg
- Empagliflozin 25 mg (Drug Naive): Patients rolled over from trial 1245.20
  Empagliflozin 25 mg tablets once daily
  Placebo: Placebo matching Sitagliptin
  Placebo: Placebo matching Empagliflozin 10 mg
- Placebo (Drug Naive): Patients rolled over from trial 1245.20
  Placebo tablets matching Empagliflozin / Sitagliptin once daily
  Placebo: Placebo matching Empagliflozin 10 mg
  Placebo: Placebo matching Sitagliptin
  Placebo: Placebo matching Empagliflozin 25 mg
- Sitagliptin 100mg (Drug Naive): Patients rolled over from trial 1245.20
  Sitagliptin once daily
  Placebo: Placebo matching Empagliflozin 25 mg
  Placebo: Placebo matching Empagliflozin 10 mg
  Sitagliptin 100mg: Sitagliptin once daily
- Empagliflozin 10 mg (Pioglitazone): Patients rolled over from trial 1245.19
  Empagliflozin 10 mg tablets once daily
  Empagliflozin 10 mg: Empagliflozin 10 mg tablets once daily
  Placebo: Placebo matching Empagliflozin 25 mg
- Empagliflozin 25 mg (Pioglitazone): Patients rolled over from trial 1245.19
  Empagliflozin 25 mg tablets once daily
  Empagliflozin 25 mg: Empagliflozin 25 mg tablets once daily
  Placebo: Placebo matching Empagliflozin 10 mg
- Placebo (Pioglitazone): Patients rolled over from trial 1245.19
  Placebo tablets matching Empagliflozin once daily
  Placebo: Placebo matching Empagliflozin 10 mg
  Placebo: Placebo matching Empagliflozin 25 mg
- Empagliflozin 10 mg (Metformin): Patients rolled over from trial 1245.23
  Empagliflozin 10 mg tablets once daily
  Placebo: Placebo matching Empagliflozin 25 mg
  Empagliflozin 10 mg: Empagliflozin 10 mg once daily
- Empagliflozin 25 mg (Metformin); Empagliflozin 25 mg (Metformin+Sulfonylurea): Patients rolled over from trial 1245.23
  Empagliflozin 25 mg tablets once daily
  Empagliflozin 25 mg: Empagliflozin 25 mg tablets once daily
  Placebo: Placebo matching Empagliflozin 10 mg
- Placebo (Metformin): Patients rolled over from trial 1245.23
  Placebo tablets matching Empagliflozin once daily
  Placebo: Placebo matching Empagliflozin 10 mg
  Placebo: Placebo matching Empagliflozin 25 mg
- Empagliflozin 10 mg (Metformin+Sulfonylurea): Patients rolled over from trial 1245.23
  Empagliflozin 10 mg tablets once daily
  Empagliflozin 10 mg: Empagliflozin 10 mg tablets once daily
  Placebo: Placebo matching Empagliflozin 25 mg
- Placebo (Metformin+Sulfonylurea): Patients rolled over from trial 1245.23
  Placebo tablets matching Empagliflozin
  Placebo: Placebo matching Empagliflozin 10 mg
  Placebo: Placebo matching Empagliflozin 25 mg
Period: Overall Study
Arm/Group | Empagliflozin 10 mg (Drug Naive) | Empagliflozin 25 mg (Drug Naive) | Placebo (Drug Naive) | Sitagliptin 100mg (Drug Naive) | Empagliflozin 10 mg (Pioglitazone) | Empagliflozin 25 mg (Pioglitazone) | Placebo (Pioglitazone) | Empagliflozin 10 mg (Metformin) | Empagliflozin 25 mg (Metformin) | Placebo (Metformin) | Empagliflozin 10 mg (Metformin+Sulfonylurea) | Empagliflozin 25 mg (Metformin+Sulfonylurea) | Placebo (Metformin+Sulfonylurea)
Started | 224 | 224 | 228 | 223 | 165 | 168 | 166 | 217 | 214 | 207 | 226 | 218 | 225
Completed | 147 | 143 | 119 | 136 | 93 | 94 | 78 | 162 | 139 | 121 | 150 | 150 | 127
Not Completed | 77 | 81 | 109 | 87 | 72 | 74 | 88 | 55 | 75 | 86 | 76 | 68 | 98
Not completed — Death | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 3 | 2 | 5 | 5 | 3 | 4 | 2 | 2 | 1 | 4 | 2 | 1 | 2
Not completed — Withdrawal by Subject | 15 | 14 | 12 | 13 | 8 | 7 | 13 | 9 | 12 | 13 | 11 | 13 | 16
Not completed — discontinued in preceding trial | 18 | 20 | 41 | 17 | 11 | 12 | 18 | 8 | 17 | 21 | 17 | 17 | 24
Not completed — did not continue in extension | 41 | 45 | 51 | 51 | 48 | 50 | 54 | 36 | 44 | 48 | 45 | 34 | 56
Not completed — Not treated | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 2 | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS): which contained all randomised patients who received at least 1 dose of study drug and had a baseline HbA1c assessment, irrespective of participation in the extension trial.
Groups:
- Empagliflozin 10 mg (Drug Naive): Patients rolled over from trial 1245.20
  Empagliflozin 10 mg tablets once daily
  Empagliflozin 10 mg: Empagliflozin 10 mg tablets once daily
  Placebo: Placebo matching Sitagliptin
  Placebo: Placebo matching Empagliflozin 25 mg
- Empagliflozin 25 mg (Drug Naive): Patients rolled over from trial 1245.20
  Empagliflozin 25 mg tablets once daily
  Placebo: Placebo matching Sitagliptin
  Empagliflozin 25 mg: Empagliflozin 25 mg tablets once daily
  Placebo: Placebo matching Empagliflozin 10 mg
- Sitagliptin 100 mg (Drug Naive): Patients rolled over from trial 1245.20
  Sitagliptin once daily
  Placebo: Placebo matching Empagliflozin 25 mg
  Placebo: Placebo matching Empagliflozin 10 mg
  Sitagliptin 100 mg: Sitagliptin once daily
- Total: Total of all reporting groups
Arm/Group | Empagliflozin 10 mg (Drug Naive) | Empagliflozin 25 mg (Drug Naive) | Placebo (Drug Naive) | Sitagliptin 100 mg (Drug Naive) | Empagliflozin 10 mg (Pioglitazone) | Empagliflozin 25 mg (Pioglitazone) | Placebo (Pioglitazone) | Empagliflozin 10 mg (Metformin) | Empagliflozin 25 mg (Metformin) | Placebo (Metformin) | Empagliflozin 10 mg (Metformin+Sulfonylurea) | Empagliflozin 25 mg (Metformin+Sulfonylurea) | Placebo (Metformin+Sulfonylurea) | Total
Number analyzed (Participants) | 224 | 224 | 228 | 223 | 165 | 168 | 165 | 217 | 213 | 207 | 225 | 216 | 225 | 2700
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.2 (11.6) | 53.8 (11.6) | 54.9 (10.9) | 55.1 (9.9) | 54.7 (9.9) | 54.2 (8.9) | 54.6 (10.5) | 55.5 (9.9) | 55.6 (10.2) | 56.0 (9.7) | 57.0 (9.2) | 57.4 (9.3) | 56.9 (9.2) | 55.6 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 82 | 79 | 105 | 82 | 82 | 83 | 92 | 92 | 93 | 91 | 112 | 102 | 113 | 1208
  Male | 142 | 145 | 123 | 141 | 83 | 85 | 73 | 125 | 120 | 116 | 113 | 114 | 112 | 1492

OUTCOME MEASURES:

1. Primary Outcome: Changes From Baseline in Glycosylated Haemoglobin (HbA1c) (%) After 52 Weeks of Treatment
Description: Change from baseline in HbA1c after 52 weeks
Time Frame: Baseline and 52 weeks
Population: Full Analysis Set (FAS) which contained all randomised patients who received at least 1 dose of study drug and had a baseline HbA1c assessment, irrespective of participation in the extension trial.
  (LOCF:Last observation carried forward)
Measure: Least Squares Mean (Standard Error); unit: % of HbA1c
Groups:
- BI 10773 Low (Drug Naive): Patients rolled over from trial 1245.20
  BI 10773 tablets once daily
  BI 10773: BI 10773 tablets once daily
  Placebo: Placebo matching Sitagliptin
  Placebo: Placebo matching BI 10773 high dose
- BI 10773 High (Drug Naive): Patients rolled over from trial 1245.20
  BI 10773 tablets once daily
  Placebo: Placebo matching Sitagliptin
  BI 10773: BI 10773 tablets once daily
  Placebo: Placebo matching BI 10773 low dose
- Placebo (Drug Naive): Patients rolled over from trial 1245.20
  Placebo tablets matching BI 10773 / Sitagliptin once daily
  Placebo: Placebo matching BI 10773 low dose
  Placebo: Placebo matching Sitagliptin
  Placebo: Placebo matching BI 10773 high dose
- Sitagliptin 100mg (Drug Naive): Patients rolled over from trial 1245.20
  Sitagliptin once daily
  Placebo: Placebo matching BI 10773 high dose
  Placebo: Placebo matching BI 10773 low dose
  Sitagliptin 100mg: Sitagliptin once daily
- BI 10773 Low (Pioglitazone): Patients rolled over from trial 1245.19
  BI 10773 tablets once daily
  BI 10773: BI 10773 tablets once daily
  Placebo: Placebo matching BI 10773 high dose
- BI 10773 High (Pioglitazone): Patients rolled over from trial 1245.19
  BI 10773 tablets once daily
  BI 10773: BI 10773 tablets once daily
  Placebo: Placebo matching BI 10773 low dose
- Placebo (Pioglitazone): Patients rolled over from trial 1245.19
  Placebo tablets matching BI 10773 once daily
  Placebo: Placebo matching BI 10773 low dose
  Placebo: Placebo matching BI 10773 high dose
- BI 10773 Low (Metformin): Patients rolled over from trial 1245.23
  BI 10773 tablets once daily
  Placebo: Placebo matching BI 10773 high dose
  BI 10773: BI 10773 tablets once daily
- BI 10773 High (Metformin); BI 10773 High (Metformin+Sulfonylurea): Patients rolled over from trial 1245.23
  BI 10773 tablets once daily
  BI 10773: BI 10773 tablets once daily
  Placebo: Placebo matching BI 10773 low dose
- Placebo (Metformin): Patients rolled over from trial 1245.23
  Placebo tablets matching BI 10773 once daily
  Placebo: Placebo matching BI 10773 low dose
  Placebo: Placebo matching BI 10773 high dose
- BI 10773 Low (Metformin+Sulfonylurea): Patients rolled over from trial 1245.23
  BI 10773 tablets once daily
  BI 10773: BI 10773 tablets once daily
  Placebo: Placebo matching BI 10773 high dose
- Placebo (Metformin+Sulfonylurea): Patients rolled over from trial 1245.23
  Placebo tablets matching BI 10773
  Placebo: Placebo matching BI 10773 low dose
  Placebo: Placebo matching BI 10773 high dose
Arm/Group | BI 10773 Low (Drug Naive) | BI 10773 High (Drug Naive) | Placebo (Drug Naive) | Sitagliptin 100mg (Drug Naive) | BI 10773 Low (Pioglitazone) | BI 10773 High (Pioglitazone) | Placebo (Pioglitazone) | BI 10773 Low (Metformin) | BI 10773 High (Metformin) | Placebo (Metformin) | BI 10773 Low (Metformin+Sulfonylurea) | BI 10773 High (Metformin+Sulfonylurea) | Placebo (Metformin+Sulfonylurea)
Number analyzed (Participants) | 224 | 224 | 228 | 223 | 165 | 168 | 165 | 217 | 213 | 207 | 225 | 216 | 225
% of HbA1c | -0.70 (0.05) | -0.82 (0.05) | 0.09 (0.05) | -0.58 (0.05) | -0.63 (0.07) | -0.71 (0.07) | -0.03 (0.07) | -0.69 (0.05) | -0.76 (0.05) | -0.07 (0.05) | -0.78 (0.05) | -0.74 (0.05) | -0.04 (0.05)
Statistical Analysis 1: Comparison: BI 10773 Low (Drug Naive) vs Placebo (Drug Naive); statistical analysis at week 52; Test type: Superiority or Other; p < 0.0001, ANCOVA — Model includes baseline HbA1c as a linear covariate, baseline estimated glomerular filtration rate (eGFR), geographic region, and treatment as fixed effects; Adjusted mean difference = -0.79, 95% CI 2-sided [-0.94 to -0.64], Standard Error of Mean 0.08
Statistical Analysis 2: Comparison: BI 10773 High (Drug Naive) vs Placebo (Drug Naive); statistical analysis at week 52; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Adjusted mean difference = -0.91, 95% CI 2-sided [-1.06 to -0.76], Standard Error of Mean 0.08
Statistical Analysis 3: Comparison: Placebo (Drug Naive) vs Sitagliptin 100mg (Drug Naive); statistical analysis at week 52; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Adjusted mean difference = -0.67, 95% CI 2-sided [-0.82 to -0.52], Standard Error of Mean 0.08
Statistical Analysis 4: Comparison: BI 10773 Low (Drug Naive) vs Sitagliptin 100mg (Drug Naive); statistical analysis at week 52; Test type: Superiority or Other; p = 0.1245, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Adjusted mean difference = -0.12, 95% CI 2-sided [-0.27 to 0.03], Standard Error of Mean 0.08
Statistical Analysis 5: Comparison: BI 10773 High (Drug Naive) vs Sitagliptin 100mg (Drug Naive); statistical analysis at week 52; Test type: Superiority or Other; p = 0.0022, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Adjusted mean difference = -0.24, 95% CI 2-sided [-0.39 to -0.09], Standard Error of Mean 0.08
Statistical Analysis 6: Comparison: BI 10773 Low (Pioglitazone) vs Placebo (Pioglitazone); Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Adjusted mean difference = -0.60, 95% CI 2-sided [-0.79 to -0.41], Standard Error of Mean 0.10
Statistical Analysis 7: Comparison: BI 10773 High (Pioglitazone) vs Placebo (Pioglitazone); Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Adjusted mean difference = -0.68, 95% CI 2-sided [-0.87 to -0.49], Standard Error of Mean 0.10
Statistical Analysis 8: Comparison: BI 10773 Low (Metformin) vs Placebo (Metformin); Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Adjusted mean difference = -0.62, 95% CI 2-sided [-0.75 to -0.48], Standard Error of Mean 0.07
Statistical Analysis 9: Comparison: BI 10773 High (Metformin) vs Placebo (Metformin); Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Adjusted mean difference = -0.69, 95% CI 2-sided [-0.83 to -0.55], Standard Error of Mean 0.07
Statistical Analysis 10: Comparison: BI 10773 Low (Metformin+Sulfonylurea) vs Placebo (Metformin+Sulfonylurea); Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Adjusted mean difference = -0.74, 95% CI 2-sided [-0.89 to -0.59], Standard Error of Mean 0.08
Statistical Analysis 11: Comparison: BI 10773 High (Metformin+Sulfonylurea) vs Placebo (Metformin+Sulfonylurea); Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Adjusted mean difference = -0.70, 95% CI 2-sided [-0.85 to -0.55], Standard Error of Mean 0.08

2. Secondary Outcome: HbA1c (%) Changes From Baseline After 76 Weeks of Treatment
Description: Change from baseline in HbA1c (%) after 76 weeks using MMRM approach
Time Frame: Baseline and 76 weeks
Population: Full Analysis Set (FAS) which contained all randomised patients who received at least 1 dose of study drug and had a baseline HbA1c assessment, irrespective of participation in the extension trial. (OC: Observed cases)
Measure: Least Squares Mean (Standard Error); unit: % of HbA1c
Arm/Group | BI 10773 Low (Drug Naive) | BI 10773 High (Drug Naive) | Placebo (Drug Naive) | Sitagliptin 100mg (Drug Naive) | BI 10773 Low (Pioglitazone) | BI 10773 High (Pioglitazone) | Placebo (Pioglitazone) | BI 10773 Low (Metformin) | BI 10773 High (Metformin) | Placebo (Metformin) | BI 10773 Low (Metformin+Sulfonylurea) | BI 10773 High (Metformin+Sulfonylurea) | Placebo (Metformin+Sulfonylurea)
Number analyzed (Participants) | 132 | 132 | 65 | 108 | 71 | 78 | 31 | 130 | 118 | 70 | 110 | 103 | 76
% of HbA1c | -0.70 (0.07) | -0.77 (0.07) | 0.13 (0.08) | -0.48 (0.07) | -0.67 (0.09) | -0.77 (0.08) | -0.05 (0.12) | -0.60 (0.06) | -0.76 (0.07) | 0.07 (0.08) | -0.75 (0.08) | -0.75 (0.08) | 0.06 (0.09)
Statistical Analysis 1: Comparison: BI 10773 Low (Drug Naive) vs Placebo (Drug Naive); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Model includes baseline HbA1c as a covariate, baseline estimated glomerular filtration rate (eGFR), geographic region, visit, treatment as fixed effects, and visit by treatment interaction; Adjusted mean difference = -0.82, 95% CI 2-sided [-1.04 to -0.61], Standard Error of Mean 0.11
Statistical Analysis 2: Comparison: BI 10773 High (Drug Naive) vs Placebo (Drug Naive); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]; Adjusted mean difference = -0.90, 95% CI 2-sided [-1.11 to -0.69], Standard Error of Mean 0.11
Statistical Analysis 3: Comparison: BI 10773 Low (Drug Naive) vs Sitagliptin 100mg (Drug Naive); Test type: Superiority or Other; p = 0.0322, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]; Adjusted mean difference = -0.21, 95% CI 2-sided [-0.41 to -0.02], Standard Error of Mean 0.10
Statistical Analysis 4: Comparison: BI 10773 High (Drug Naive) vs Sitagliptin 100mg (Drug Naive); Test type: Superiority or Other; p = 0.0038, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]; Adjusted mean difference = -0.29, 95% CI 2-sided [-0.48 to -0.09], Standard Error of Mean 0.10
Statistical Analysis 5: Comparison: Placebo (Drug Naive) vs Sitagliptin 100mg (Drug Naive); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]; Adjusted mean difference = -0.61, 95% CI 2-sided [-0.83 to -0.40], Standard Error of Mean 0.11
Statistical Analysis 6: Comparison: BI 10773 Low (Pioglitazone) vs Placebo (Pioglitazone); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]; Adjusted mean difference = -0.62, 95% CI 2-sided [-0.90 to -0.33], Standard Error of Mean 0.15
Statistical Analysis 7: Comparison: BI 10773 High (Pioglitazone) vs Placebo (Pioglitazone); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]; Adjusted mean difference = -0.72, 95% CI 2-sided [-1.00 to -0.44], Standard Error of Mean 0.14
Statistical Analysis 8: Comparison: BI 10773 Low (Metformin) vs Placebo (Metformin); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]; Adjusted mean difference = -0.67, 95% CI 2-sided [-0.87 to -0.47], Standard Error of Mean 0.10
Statistical Analysis 9: Comparison: BI 10773 High (Metformin) vs Placebo (Metformin); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]; Adjusted mean difference = -0.83, 95% CI 2-sided [-1.04 to -0.63], Standard Error of Mean 0.10
Statistical Analysis 10: Comparison: BI 10773 Low (Metformin+Sulfonylurea) vs Placebo (Metformin+Sulfonylurea); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]; Adjusted mean difference = -0.80, 95% CI 2-sided [-1.04 to -0.57], Standard Error of Mean 0.12
Statistical Analysis 11: Comparison: BI 10773 High (Metformin+Sulfonylurea) vs Placebo (Metformin+Sulfonylurea); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]; Adjusted mean difference = -0.80, 95% CI 2-sided [-1.04 to -0.56], Standard Error of Mean 0.12

3. Secondary Outcome: Systolic Blood Pressure: Change From Baseline After 52 Weeks of Treatment
Description: Systolic blood pressure - change from baseline after 52 weeks of treatment
Time Frame: Baseline and 52 weeks
Population: Full Analysis Set (FAS) which contained all randomised patients who received at least 1 dose of study drug and had a baseline systolic blood pressure assessment, irrespective of participation in the extension trial. (LOCF)
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | BI 10773 Low (Drug Naive) | BI 10773 High (Drug Naive) | Placebo (Drug Naive) | Sitagliptin 100mg (Drug Naive) | BI 10773 Low (Pioglitazone) | BI 10773 High (Pioglitazone) | Placebo (Pioglitazone) | BI 10773 Low (Metformin) | BI 10773 High (Metformin) | Placebo (Metformin) | BI 10773 Low (Metformin+Sulfonylurea) | BI 10773 High (Metformin+Sulfonylurea) | Placebo (Metformin+Sulfonylurea)
Number analyzed (Participants) | 224 | 224 | 228 | 223 | 165 | 168 | 165 | 217 | 213 | 207 | 225 | 216 | 225
mmHg | -4.9 (0.8) | -4.5 (0.8) | -1.6 (0.8) | -0.2 (0.8) | -1.8 (0.9) | -3.3 (0.9) | 0.6 (0.9) | -3.6 (0.7) | -5.2 (0.7) | -0.7 (0.7) | -3.1 (0.7) | -2.7 (0.7) | -0.2 (0.7)
Statistical Analysis 1: Comparison: BI 10773 Low (Drug Naive) vs Placebo (Drug Naive); Test type: Superiority or Other; p < 0.0001, ANCOVA — Model includes baseline sys blood pressure, baseline HbA1c as covariates, baseline eGFR, geographic region, and treatment as fixed effects; Adjusted mean difference = -4.6, 95% CI 2-sided [-6.8 to -2.5], Standard Error of Mean 1.1
Statistical Analysis 2: Comparison: BI 10773 High (Drug Naive) vs Placebo (Drug Naive); Test type: Superiority or Other; p = 0.0001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Adjusted mean difference = -4.2, 95% CI 2-sided [-6.4 to -2.1], Standard Error of Mean 1.1
Statistical Analysis 3: Comparison: Placebo (Drug Naive) vs Sitagliptin 100mg (Drug Naive); Test type: Superiority or Other; p = 0.2107, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Adjusted mean difference = -1.4, 95% CI 2-sided [-3.5 to 0.8], Standard Error of Mean 1.1
Statistical Analysis 4: Comparison: BI 10773 Low (Drug Naive) vs Sitagliptin 100mg (Drug Naive); Test type: Superiority or Other; p = 0.0033, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Adjusted mean difference = -3.3, 95% CI 2-sided [-5.4 to -1.1], Standard Error of Mean 1.1
Statistical Analysis 5: Comparison: BI 10773 High (Drug Naive) vs Sitagliptin 100mg (Drug Naive); Test type: Superiority or Other; p = 0.0105, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Adjusted mean difference = -2.8, 95% CI 2-sided [-5.0 to -0.7], Standard Error of Mean 1.1
Statistical Analysis 6: Comparison: BI 10773 Low (Pioglitazone) vs Placebo (Pioglitazone); Test type: Superiority or Other; p = 0.0543, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Adjusted mean difference = -2.4, 95% CI 2-sided [-4.9 to 0.0], Standard Error of Mean 1.3
Statistical Analysis 7: Comparison: BI 10773 High (Pioglitazone) vs Placebo (Pioglitazone); Test type: Superiority or Other; p = 0.0019, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Adjusted mean difference = -3.9, 95% CI 2-sided [-6.4 to -1.5], Standard Error of Mean 1.2
Statistical Analysis 8: Comparison: BI 10773 Low (Metformin) vs Placebo (Metformin); Test type: Superiority or Other; p = 0.0045, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Adjusted mean difference = -3.0, 95% CI 2-sided [-5.0 to -0.9], Standard Error of Mean 1.0
Statistical Analysis 9: Comparison: BI 10773 High (Metformin) vs Placebo (Metformin); Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Adjusted mean difference = -4.5, 95% CI 2-sided [-6.6 to -2.5], Standard Error of Mean 1.0
Statistical Analysis 10: Comparison: BI 10773 Low (Metformin+Sulfonylurea) vs Placebo (Metformin+Sulfonylurea); Test type: Superiority or Other; p = 0.0031, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Adjusted mean difference = -2.9, 95% CI 2-sided [-4.8 to -1.0], Standard Error of Mean 1.0
Statistical Analysis 11: Comparison: BI 10773 High (Metformin+Sulfonylurea) vs Placebo (Metformin+Sulfonylurea); Test type: Superiority or Other; p = 0.0096, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Adjusted mean difference = -2.5, 95% CI 2-sided [-4.4 to -0.6], Standard Error of Mean 1.0

4. Primary Outcome: Changes From Baseline in HbA1c (%) After 76 Weeks of Treatment
Description: Change from baseline in HbA1c after 76 weeks
Time Frame: Baseline and 76 weeks
Population: Full Analysis Set (FAS) which contained all randomised patients who received at least 1 dose of study drug and had a baseline HbA1c assessment, irrespective of participation in the extension trial. (LOCF)
Measure: Least Squares Mean (Standard Deviation); unit: % of HbA1c
Arm/Group | BI 10773 Low (Drug Naive) | BI 10773 High (Drug Naive) | Placebo (Drug Naive) | Sitagliptin 100mg (Drug Naive) | BI 10773 Low (Pioglitazone) | BI 10773 High (Pioglitazone) | Placebo (Pioglitazone) | BI 10773 Low (Metformin) | BI 10773 High (Metformin) | Placebo (Metformin) | BI 10773 Low (Metformin+Sulfonylurea) | BI 10773 High (Metformin+Sulfonylurea) | Placebo (Metformin+Sulfonylurea)
Number analyzed (Participants) | 224 | 224 | 228 | 223 | 165 | 168 | 165 | 217 | 213 | 207 | 225 | 216 | 225
% of HbA1c | -0.65 (0.06) | -0.76 (0.06) | 0.13 (0.06) | -0.53 (0.06) | -0.61 (0.07) | -0.70 (0.07) | -0.01 (0.07) | -0.62 (0.05) | -0.74 (0.05) | -0.01 (0.05) | -0.74 (0.06) | -0.72 (0.06) | -0.03 (0.06)
Statistical Analysis 1: Comparison: BI 10773 Low (Drug Naive) vs Placebo (Drug Naive); Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Adjusted mean difference = -0.78, 95% CI 2-sided [-0.94 to -0.63], Standard Error of Mean 0.08
Statistical Analysis 2: Comparison: BI 10773 High (Drug Naive) vs Placebo (Drug Naive); Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Adjusted mean difference = -0.89, 95% CI 2-sided [-1.04 to -0.73], Standard Error of Mean 0.08
Statistical Analysis 3: Comparison: Placebo (Drug Naive) vs Sitagliptin 100mg (Drug Naive); Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Adjusted mean difference = -0.66, 95% CI 2-sided [-0.82 to -0.51], Standard Error of Mean 0.08
Statistical Analysis 4: Comparison: BI 10773 Low (Drug Naive) vs Sitagliptin 100mg (Drug Naive); Test type: Superiority or Other; p = 0.1310, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Adjusted mean difference = -0.12, 95% CI 2-sided [-0.28 to 0.04], Standard Error of Mean 0.08
Statistical Analysis 5: Comparison: BI 10773 High (Drug Naive) vs Sitagliptin 100mg (Drug Naive); Test type: Superiority or Other; p = 0.0050, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Adjusted mean difference = -0.22, 95% CI 2-sided [-0.38 to -0.07], Standard Error of Mean 0.08
Statistical Analysis 6: Comparison: BI 10773 Low (Pioglitazone) vs Placebo (Pioglitazone); Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Adjusted mean difference = -0.59, 95% CI 2-sided [-0.79 to -0.40], Standard Error of Mean 0.10
Statistical Analysis 7: Comparison: BI 10773 High (Pioglitazone) vs Placebo (Pioglitazone); Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Adjusted mean difference = -0.69, 95% CI 2-sided [-0.88 to -0.50], Standard Error of Mean 0.10
Statistical Analysis 8: Comparison: BI 10773 Low (Metformin) vs Placebo (Metformin); Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Adjusted mean difference = -0.61, 95% CI 2-sided [-0.75 to -0.46], Standard Error of Mean 0.07
Statistical Analysis 9: Comparison: BI 10773 High (Metformin) vs Placebo (Metformin); Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Adjusted mean difference = -0.73, 95% CI 2-sided [-0.88 to -0.58], Standard Error of Mean 0.07
Statistical Analysis 10: Comparison: BI 10773 Low (Metformin+Sulfonylurea) vs Placebo (Metformin+Sulfonylurea); Test type: Superiority or Other; p < 0.0001, ANCOVA; Adjusted mean difference = -0.72, 95% CI 2-sided [-0.87 to -0.56], Standard Error of Mean 0.08
Statistical Analysis 11: Comparison: BI 10773 High (Metformin+Sulfonylurea) vs Placebo (Metformin+Sulfonylurea); Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Adjusted mean difference = -0.69, 95% CI 2-sided [-0.85 to -0.53], Standard Error of Mean 0.08

5. Secondary Outcome: Systolic Blood Pressure: Change From Baseline After 76 Weeks of Treatment
Description: Systolic blood pressure - change from baseline after 76 weeks of treatment
Time Frame: Baseline and 76 weeks
Population: Full Analysis Set (FAS) which contained all randomised patients who received at least 1 dose of study drug and had a baseline systolic blood pressure assessment, irrespective of participation in the extension trial -LOCF
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | BI 10773 Low (Drug Naive) | BI 10773 High (Drug Naive) | Placebo (Drug Naive) | Sitagliptin 100mg (Drug Naive) | BI 10773 Low (Pioglitazone) | BI 10773 High (Pioglitazone) | Placebo (Pioglitazone) | BI 10773 Low (Metformin) | BI 10773 High (Metformin) | Placebo (Metformin) | BI 10773 Low (Metformin+Sulfonylurea) | BI 10773 High (Metformin+Sulfonylurea) | Placebo (Metformin+Sulfonylurea)
Number analyzed (Participants) | 224 | 224 | 228 | 223 | 165 | 168 | 165 | 217 | 213 | 207 | 225 | 216 | 225
mmHg | -4.1 (0.8) | -4.2 (0.8) | -0.7 (0.8) | -0.3 (0.8) | -1.7 (0.9) | -3.4 (0.9) | 0.3 (0.9) | -5.2 (0.8) | -4.5 (0.8) | -0.8 (0.8) | -3.8 (0.7) | -3.7 (0.7) | -1.6 (0.7)
Statistical Analysis 1: Comparison: BI 10773 Low (Drug Naive) vs Placebo (Drug Naive); Test type: Superiority or Other; p = 0.0025, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Adjusted mean difference = -3.4, 95% CI 2-sided [-5.5 to -1.2], Standard Error of Mean 1.1
Statistical Analysis 2: Comparison: BI 10773 High (Drug Naive) vs Placebo (Drug Naive); Test type: Superiority or Other; p = 0.0021, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Adjusted mean difference = -3.4, 95% CI 2-sided [-5.6 to -1.2], Standard Error of Mean 1.1
Statistical Analysis 3: Comparison: Placebo (Drug Naive) vs Sitagliptin 100mg (Drug Naive); Test type: Superiority or Other; p = 0.7241, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Adjusted mean difference = 0.4, 95% CI 2-sided [-1.8 to 2.6], Standard Error of Mean 1.1
Statistical Analysis 4: Comparison: BI 10773 Low (Drug Naive) vs Sitagliptin 100mg (Drug Naive); Test type: Superiority or Other; p = 0.0008, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Adjusted mean difference = -3.7, 95% CI 2-sided [-5.9 to -1.6], Standard Error of Mean 1.1
Statistical Analysis 5: Comparison: BI 10773 High (Drug Naive) vs Sitagliptin 100mg (Drug Naive); Test type: Superiority or Other; p = 0.0007, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Adjusted mean difference = -3.8, 95% CI 2-sided [-6.0 to -1.6], Standard Error of Mean 1.1
Statistical Analysis 6: Comparison: BI 10773 Low (Pioglitazone) vs Placebo (Pioglitazone); Test type: Superiority or Other; p = 0.0987, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Adjusted mean difference = -2.0, 95% CI 2-sided [-4.5 to 0.4], Standard Error of Mean 1.2
Statistical Analysis 7: Comparison: BI 10773 High (Pioglitazone) vs Placebo (Pioglitazone); Test type: Superiority or Other; p = 0.0028, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Adjusted mean difference = -3.7, 95% CI 2-sided [-6.1 to -1.3], Standard Error of Mean 1.2
Statistical Analysis 8: Comparison: BI 10773 Low (Metformin) vs Placebo (Metformin); Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Adjusted mean difference = -4.4, 95% CI 2-sided [-6.6 to -2.3], Standard Error of Mean 1.1
Statistical Analysis 9: Comparison: BI 10773 High (Metformin) vs Placebo (Metformin); Test type: Superiority or Other; p = 0.0008, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Adjusted mean difference = -3.7, 95% CI 2-sided [-5.9 to -1.5], Standard Error of Mean 1.1
Statistical Analysis 10: Comparison: BI 10773 Low (Metformin+Sulfonylurea) vs Placebo (Metformin+Sulfonylurea); Test type: Superiority or Other; p = 0.0213, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Adjusted mean difference = -2.2, 95% CI 2-sided [-4.1 to -0.3], Standard Error of Mean 1.0
Statistical Analysis 11: Comparison: BI 10773 High (Metformin+Sulfonylurea) vs Placebo (Metformin+Sulfonylurea); Test type: Superiority or Other; p = 0.0288, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Adjusted mean difference = -2.1, 95% CI 2-sided [-4.1 to -0.2], Standard Error of Mean 1.0

6. Secondary Outcome: Diastolic Blood Pressure: Change From Baseline After 52 Weeks of Treatment
Description: Diastolic blood pressure - change from baseline after 52 weeks of treatment
Time Frame: Baseline and 52 weeks
Population: Full Analysis Set (FAS) which contained all randomised patients who received at least 1 dose of study drug and had a baseline diastolic blood pressure assessment, irrespective of participation in the extension trial -LOCF
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | BI 10773 Low (Drug Naive) | BI 10773 High (Drug Naive) | Placebo (Drug Naive) | Sitagliptin 100mg (Drug Naive) | BI 10773 Low (Pioglitazone) | BI 10773 High (Pioglitazone) | Placebo (Pioglitazone) | BI 10773 Low (Metformin) | BI 10773 High (Metformin) | Placebo (Metformin) | BI 10773 Low (Metformin+Sulfonylurea) | BI 10773 High (Metformin+Sulfonylurea) | Placebo (Metformin+Sulfonylurea)
Number analyzed (Participants) | 224 | 224 | 228 | 223 | 165 | 168 | 165 | 217 | 213 | 207 | 225 | 216 | 225
mmHg | -1.3 (0.5) | -1.9 (0.5) | -0.2 (0.5) | -0.3 (0.5) | -1.6 (0.5) | -2.2 (0.5) | 0.4 (0.5) | -2.2 (0.5) | -2.1 (0.5) | -0.4 (0.5) | -1.7 (0.5) | -1.6 (0.5) | -1.0 (0.5)
Statistical Analysis 1: Comparison: BI 10773 Low (Drug Naive) vs Placebo (Drug Naive); Test type: Superiority or Other; p = 0.1058, ANCOVA — Model includes baseline diastolic blood pressure, baseline HbA1c as covariates, baseline eGFR, geographic region, and treatment as fixed effects; Adjusted mean difference = -1.1, 95% CI 2-sided [-2.4 to 0.2], Standard Error of Mean 0.7
Statistical Analysis 2: Comparison: BI 10773 High (Drug Naive) vs Placebo (Drug Naive); Test type: Superiority or Other; p = 0.0109, ANCOVA — [p-value comment as in outcome 6, analysis 1]; Adjusted mean difference = -1.7, 95% CI 2-sided [-3.1 to -0.4], Standard Error of Mean 0.7
Statistical Analysis 3: Comparison: Placebo (Drug Naive) vs Sitagliptin 100mg (Drug Naive); Test type: Superiority or Other; p = 0.8259, ANCOVA — [p-value comment as in outcome 6, analysis 1]; Adjusted mean difference = -0.2, 95% CI 2-sided [-1.5 to 1.2], Standard Error of Mean 0.7
Statistical Analysis 4: Comparison: BI 10773 Low (Drug Naive) vs Sitagliptin 100mg (Drug Naive); Test type: Superiority or Other; p = 0.1660, ANCOVA — [p-value comment as in outcome 6, analysis 1]; Adjusted mean difference = -0.9, 95% CI 2-sided [-2.3 to 0.4], Standard Error of Mean 0.7
Statistical Analysis 5: Comparison: BI 10773 High (Drug Naive) vs Sitagliptin 100mg (Drug Naive); Test type: Superiority or Other; p = 0.0212, ANCOVA — [p-value comment as in outcome 6, analysis 1]; Adjusted mean difference = -1.6, 95% CI 2-sided [-2.9 to -0.2], Standard Error of Mean 0.7
Statistical Analysis 6: Comparison: BI 10773 Low (Pioglitazone) vs Placebo (Pioglitazone); Test type: Superiority or Other; p = 0.0076, ANCOVA — [p-value comment as in outcome 6, analysis 1]; Adjusted mean difference = -2.0, 95% CI 2-sided [-3.4 to -0.5], Standard Error of Mean 0.7
Statistical Analysis 7: Comparison: BI 10773 High (Pioglitazone) vs Placebo (Pioglitazone); Test type: Superiority or Other; p = 0.0003, ANCOVA — [p-value comment as in outcome 6, analysis 1]; Adjusted mean difference = -2.6, 95% CI 2-sided [-4.1 to -1.2], Standard Error of Mean 0.7
Statistical Analysis 8: Comparison: BI 10773 Low (Metformin) vs Placebo (Metformin); Test type: Superiority or Other; p = 0.0170, ANCOVA — [p-value comment as in outcome 6, analysis 1]; Adjusted mean difference = -1.8, 95% CI 2-sided [-3.2 to -0.3], Standard Error of Mean 0.7
Statistical Analysis 9: Comparison: BI 10773 High (Metformin) vs Placebo (Metformin); Test type: Superiority or Other; p = 0.0236, ANCOVA — [p-value comment as in outcome 6, analysis 1]; Adjusted mean difference = -1.7, 95% CI 2-sided [-3.1 to -0.2], Standard Error of Mean 0.7
Statistical Analysis 10: Comparison: BI 10773 Low (Metformin+Sulfonylurea) vs Placebo (Metformin+Sulfonylurea); Test type: Superiority or Other; p = 0.2523, ANCOVA — [p-value comment as in outcome 6, analysis 1]; Adjusted mean difference = -0.7, 95% CI 2-sided [-2.0 to 0.5], Standard Error of Mean 0.6
Statistical Analysis 11: Comparison: BI 10773 High (Metformin+Sulfonylurea) vs Placebo (Metformin+Sulfonylurea); Test type: Superiority or Other; p = 0.3494, ANCOVA — [p-value comment as in outcome 6, analysis 1]; Adjusted mean difference = -0.6, 95% CI 2-sided [-1.9 to 0.7], Standard Error of Mean 0.6

7. Secondary Outcome: Diastolic Blood Pressure: Change From Baseline After 76 Weeks of Treatment
Description: Diastolic blood pressure - change from baseline after 76 weeks of treatment
Time Frame: Baseline and 76 weeks
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | BI 10773 Low (Drug Naive) | BI 10773 High (Drug Naive) | Placebo (Drug Naive) | Sitagliptin 100mg (Drug Naive) | BI 10773 Low (Pioglitazone) | BI 10773 High (Pioglitazone) | Placebo (Pioglitazone) | BI 10773 Low (Metformin) | BI 10773 High (Metformin) | Placebo (Metformin) | BI 10773 Low (Metformin+Sulfonylurea) | BI 10773 High (Metformin+Sulfonylurea) | Placebo (Metformin+Sulfonylurea)
Number analyzed (Participants) | 224 | 224 | 228 | 223 | 165 | 168 | 165 | 217 | 213 | 207 | 225 | 216 | 225
mmHg | -1.6 (0.5) | -1.6 (0.5) | -0.6 (0.5) | -0.1 (0.5) | -1.3 (0.5) | -2.0 (0.5) | 0.2 (0.5) | -2.5 (0.5) | -1.9 (0.5) | -0.5 (0.5) | -2.6 (0.5) | -2.3 (0.5) | -1.4 (0.5)
Statistical Analysis 1: Comparison: BI 10773 Low (Drug Naive) vs Placebo (Drug Naive); Test type: Superiority or Other; p = 0.1568, ANCOVA — [p-value comment as in outcome 6, analysis 1]; Adjusted mean difference = -1.0, 95% CI 2-sided [-2.3 to 0.4], Standard Error of Mean 0.7
Statistical Analysis 2: Comparison: BI 10773 High (Drug Naive) vs Placebo (Drug Naive); Test type: Superiority or Other; p = 0.1323, ANCOVA — [p-value comment as in outcome 6, analysis 1]; Adjusted mean difference = -1.0, 95% CI 2-sided [-2.4 to 0.3], Standard Error of Mean 0.7
Statistical Analysis 3: Comparison: Placebo (Drug Naive) vs Sitagliptin 100mg (Drug Naive); Test type: Superiority or Other; p = 0.4327, ANCOVA — [p-value comment as in outcome 6, analysis 1]; Adjusted mean difference = 0.5, 95% CI 2-sided [-0.8 to 1.9], Standard Error of Mean 0.7
Statistical Analysis 4: Comparison: BI 10773 Low (Drug Naive) vs Sitagliptin 100mg (Drug Naive); Test type: Superiority or Other; p = 0.0289, ANCOVA — [p-value comment as in outcome 6, analysis 1]; Adjusted mean difference = -1.5, 95% CI 2-sided [-2.8 to -0.2], Standard Error of Mean 0.7
Statistical Analysis 5: Comparison: BI 10773 High (Drug Naive) vs Sitagliptin 100mg (Drug Naive); Test type: Superiority or Other; p = 0.0231, ANCOVA — [p-value comment as in outcome 6, analysis 1]; Adjusted mean difference = -1.6, 95% CI 2-sided [-2.9 to -0.2], Standard Error of Mean 0.7
Statistical Analysis 6: Comparison: BI 10773 Low (Pioglitazone) vs Placebo (Pioglitazone); Test type: Superiority or Other; p = 0.0513, ANCOVA — [p-value comment as in outcome 6, analysis 1]; Adjusted mean difference = -1.5, 95% CI 2-sided [-3.0 to 0.0], Standard Error of Mean 0.8
Statistical Analysis 7: Comparison: BI 10773 High (Pioglitazone) vs Placebo (Pioglitazone); Test type: Superiority or Other; p = 0.0038, ANCOVA — [p-value comment as in outcome 6, analysis 1]; Adjusted mean difference = -2.2, 95% CI 2-sided [-3.7 to -0.7], Standard Error of Mean 0.8
Statistical Analysis 8: Comparison: BI 10773 Low (Metformin) vs Placebo (Metformin); Test type: Superiority or Other; p = 0.0084, ANCOVA — [p-value comment as in outcome 6, analysis 1]; Adjusted mean difference = -2.0, 95% CI 2-sided [-3.4 to -0.5], Standard Error of Mean 0.7
Statistical Analysis 9: Comparison: BI 10773 High (Metformin) vs Placebo (Metformin); Test type: Superiority or Other; p = 0.0677, ANCOVA — [p-value comment as in outcome 6, analysis 1]; Adjusted mean difference = -1.4, 95% CI 2-sided [-2.8 to 0.1], Standard Error of Mean 0.7
Statistical Analysis 10: Comparison: BI 10773 Low (Metformin+Sulfonylurea) vs Placebo (Metformin+Sulfonylurea); Test type: Superiority or Other; p = 0.0814, ANCOVA — [p-value comment as in outcome 6, analysis 1]; Adjusted mean difference = -1.1, 95% CI 2-sided [-2.4 to 0.1], Standard Error of Mean 0.7
Statistical Analysis 11: Comparison: BI 10773 High (Metformin+Sulfonylurea) vs Placebo (Metformin+Sulfonylurea); Test type: Superiority or Other; p = 0.1785, ANCOVA — [p-value comment as in outcome 6, analysis 1]; Adjusted mean difference = -0.9, 95% CI 2-sided [-2.2 to 0.4], Standard Error of Mean 0.7

8. Secondary Outcome: Body Weight (kg) Change From Baseline After 52 Weeks of Treatment
Description: Body Weight (kg) - Change From Baseline After 52 Weeks of Treatment
Time Frame: Baseline and 52 weeks
Population: Full Analysis Set (FAS) which contained all randomised patients who received at least 1 dose of study drug and had a baseline body weight assessment, irrespective of participation in the extension trial. - LOCF
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | BI 10773 Low (Drug Naive) | BI 10773 High (Drug Naive) | Placebo (Drug Naive) | Sitagliptin 100mg (Drug Naive) | BI 10773 Low (Pioglitazone) | BI 10773 High (Pioglitazone) | Placebo (Pioglitazone) | BI 10773 Low (Metformin) | BI 10773 High (Metformin) | Placebo (Metformin) | BI 10773 Low (Metformin+Sulfonylurea) | BI 10773 High (Metformin+Sulfonylurea) | Placebo (Metformin+Sulfonylurea)
Number analyzed (Participants) | 224 | 224 | 228 | 223 | 165 | 168 | 165 | 217 | 213 | 207 | 225 | 216 | 225
kg | -2.70 (0.19) | -2.61 (0.19) | -0.48 (0.19) | 0.14 (0.19) | -1.50 (0.24) | -1.40 (0.24) | 0.59 (0.24) | -2.27 (0.19) | -2.84 (0.19) | -0.54 (0.20) | -2.28 (0.18) | -2.32 (0.19) | -0.31 (0.18)
Statistical Analysis 1: Comparison: BI 10773 Low (Drug Naive) vs Placebo (Drug Naive); Test type: Superiority or Other; p < 0.0001, ANCOVA — Model includes baseline weight, baseline HbA1c as covariates, baseline eGFR, geographic region, and treatment as fixed effects; Adjusted mean difference = -2.22, 95% CI 2-sided [-2.75 to -1.69], Standard Error of Mean 0.27
Statistical Analysis 2: Comparison: BI 10773 High (Drug Naive) vs Placebo (Drug Naive); Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 8, analysis 1]; Adjusted mean difference = -2.14, 95% CI 2-sided [-2.66 to -1.61], Standard Error of Mean 0.27
Statistical Analysis 3: Comparison: Placebo (Drug Naive) vs Sitagliptin 100mg (Drug Naive); Test type: Superiority or Other; p = 0.0223, ANCOVA — [p-value comment as in outcome 8, analysis 1]; Adjusted mean difference = 0.62, 95% CI 2-sided [0.09 to 1.14], Standard Error of Mean 0.27
Statistical Analysis 4: Comparison: BI 10773 Low (Drug Naive) vs Sitagliptin 100mg (Drug Naive); Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 8, analysis 1]; Adjusted mean difference = -2.84, 95% CI 2-sided [-3.37 to -2.31], Standard Error of Mean 0.27
Statistical Analysis 5: Comparison: BI 10773 High (Drug Naive) vs Sitagliptin 100mg (Drug Naive); Test type: Superiority or Other; p < 0.0001, ANCOVA; Adjusted mean difference = -2.75, 95% CI 2-sided [-3.28 to -2.22], Standard Error of Mean 0.27
Statistical Analysis 6: Comparison: BI 10773 Low (Pioglitazone) vs Placebo (Pioglitazone); Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 8, analysis 1]; Adjusted mean difference = -2.09, 95% CI 2-sided [-2.76 to -1.41], Standard Error of Mean 0.34
Statistical Analysis 7: Comparison: BI 10773 High (Pioglitazone) vs Placebo (Pioglitazone); Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 8, analysis 1]; Adjusted mean difference = -1.99, 95% CI 2-sided [-2.66 to -1.32], Standard Error of Mean 0.34
Statistical Analysis 8: Comparison: BI 10773 Low (Metformin) vs Placebo (Metformin); Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 8, analysis 1]; Adjusted mean difference = -1.73, 95% CI 2-sided [-2.27 to -1.19], Standard Error of Mean 0.28
Statistical Analysis 9: Comparison: BI 10773 High (Metformin) vs Placebo (Metformin); Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 8, analysis 1]; Adjusted mean difference = -2.30, 95% CI 2-sided [-2.85 to -1.76], Standard Error of Mean 0.28
Statistical Analysis 10: Comparison: BI 10773 Low (Metformin+Sulfonylurea) vs Placebo (Metformin+Sulfonylurea); Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 8, analysis 1]; Adjusted mean difference = -1.97, 95% CI 2-sided [-2.48 to -1.47], Standard Error of Mean 0.26
Statistical Analysis 11: Comparison: BI 10773 High (Metformin+Sulfonylurea) vs Placebo (Metformin+Sulfonylurea); Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 8, analysis 1]; Adjusted mean difference = -2.01, 95% CI 2-sided [-2.52 to -1.50], Standard Error of Mean 0.26

9. Secondary Outcome: Body Weight (kg) Change From Baseline After 76 Weeks of Treatment
Description: Body Weight (kg) - Change From Baseline After 76 Weeks of Treatment
Time Frame: Baseline and 76 weeks
Population: Full Analysis Set (FAS) which contained all randomised patients who received at least 1 dose of study drug and had a baseline body weight assessment, irrespective of participation in the extension trial -LOCF
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | BI 10773 Low (Drug Naive) | BI 10773 High (Drug Naive) | Placebo (Drug Naive) | Sitagliptin 100mg (Drug Naive) | BI 10773 Low (Pioglitazone) | BI 10773 High (Pioglitazone) | Placebo (Pioglitazone) | BI 10773 Low (Metformin) | BI 10773 High (Metformin) | Placebo (Metformin) | BI 10773 Low (Metformin+Sulfonylurea) | BI 10773 High (Metformin+Sulfonylurea) | Placebo (Metformin+Sulfonylurea)
Number analyzed (Participants) | 224 | 224 | 228 | 223 | 165 | 168 | 165 | 217 | 213 | 207 | 225 | 216 | 225
kg | -2.24 (0.20) | -2.45 (0.20) | -0.43 (0.20) | 0.10 (0.20) | -1.47 (0.26) | -1.21 (0.26) | 0.50 (0.26) | -2.39 (0.21) | -2.65 (0.22) | -0.46 (0.22) | -2.44 (0.19) | -2.28 (0.20) | -0.63 (0.19)
Statistical Analysis 1: Comparison: BI 10773 Low (Drug Naive) vs Placebo (Drug Naive); Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 8, analysis 1]; Adjusted mean difference = -1.81, 95% CI 2-sided [-2.35 to -1.26], Standard Error of Mean 0.28
Statistical Analysis 2: Comparison: BI 10773 High (Drug Naive) vs Placebo (Drug Naive); Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 8, analysis 1]; Adjusted mean difference = -2.02, 95% CI 2-sided [-2.56 to -1.48], Standard Error of Mean 0.28
Statistical Analysis 3: Comparison: Placebo (Drug Naive) vs Sitagliptin 100mg (Drug Naive); Test type: Superiority or Other; p = 0.0546, ANCOVA — [p-value comment as in outcome 8, analysis 1]; Adjusted mean difference = 0.54, 95% CI 2-sided [-0.01 to 1.08], Standard Error of Mean 0.28
Statistical Analysis 4: Comparison: BI 10773 Low (Drug Naive) vs Sitagliptin 100mg (Drug Naive); Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 8, analysis 1]; Adjusted mean difference = -2.34, 95% CI 2-sided [-2.89 to -1.80], Standard Error of Mean 0.28
Statistical Analysis 5: Comparison: BI 10773 High (Drug Naive) vs Sitagliptin 100mg (Drug Naive); Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 8, analysis 1]; Adjusted mean difference = -2.56, 95% CI 2-sided [-3.10 to -2.01], Standard Error of Mean 0.28
Statistical Analysis 6: Comparison: BI 10773 Low (Pioglitazone) vs Placebo (Pioglitazone); Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 8, analysis 1]; Adjusted mean difference = -1.97, 95% CI 2-sided [-2.69 to -1.24], Standard Error of Mean 0.37
Statistical Analysis 7: Comparison: BI 10773 High (Pioglitazone) vs Placebo (Pioglitazone); Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 8, analysis 1]; Adjusted mean difference = -1.71, 95% CI 2-sided [-2.43 to -0.99], Standard Error of Mean 0.37
Statistical Analysis 8: Comparison: BI 10773 Low (Metformin) vs Placebo (Metformin); Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 8, analysis 1]; Adjusted mean difference = -1.93, 95% CI 2-sided [-2.52 to -1.34], Standard Error of Mean 0.30
Statistical Analysis 9: Comparison: BI 10773 High (Metformin) vs Placebo (Metformin); Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 8, analysis 1]; Adjusted mean difference = -2.19, 95% CI 2-sided [-2.79 to -1.60], Standard Error of Mean 0.30
Statistical Analysis 10: Comparison: BI 10773 Low (Metformin+Sulfonylurea) vs Placebo (Metformin+Sulfonylurea); Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 8, analysis 1]; Adjusted mean difference = -1.81, 95% CI 2-sided [-2.34 to -1.27], Standard Error of Mean 0.27
Statistical Analysis 11: Comparison: BI 10773 High (Metformin+Sulfonylurea) vs Placebo (Metformin+Sulfonylurea); Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 8, analysis 1]; Adjusted mean difference = -1.64, 95% CI 2-sided [-2.18 to -1.11], Standard Error of Mean 0.27

10. Secondary Outcome: Waist Circumference (cm) Change From Baseline After 52 Weeks of Treatment
Description: Waist circumference (cm) - change from baseline after 52 weeks of treatment
Time Frame: Baseline and 52 weeks
Population: Full Analysis Set (FAS) which contained all randomised patients who received at least 1 dose of study drug and had a baseline waist circumference assessment, irrespective of participation in the extension trial -LOCF
Measure: Least Squares Mean (Standard Error); unit: cm
Arm/Group | BI 10773 Low (Drug Naive) | BI 10773 High (Drug Naive) | Placebo (Drug Naive) | Sitagliptin 100mg (Drug Naive) | BI 10773 Low (Pioglitazone) | BI 10773 High (Pioglitazone) | Placebo (Pioglitazone) | BI 10773 Low (Metformin) | BI 10773 High (Metformin) | Placebo (Metformin) | BI 10773 Low (Metformin+Sulfonylurea) | BI 10773 High (Metformin+Sulfonylurea) | Placebo (Metformin+Sulfonylurea)
Number analyzed (Participants) | 223 | 224 | 228 | 221 | 163 | 167 | 165 | 216 | 213 | 207 | 222 | 215 | 219
cm | -2.0 (0.4) | -1.7 (0.4) | 0.1 (0.4) | 0.4 (0.4) | -1.5 (0.4) | -1.1 (0.4) | -0.1 (0.4) | -1.5 (0.3) | -2.0 (0.3) | -0.4 (0.3) | -1.5 (0.3) | -1.5 (0.3) | -0.2 (0.3)
Statistical Analysis 1: Comparison: BI 10773 Low (Drug Naive) vs Placebo (Drug Naive); Test type: Superiority or Other; p = 0.0001, ANCOVA — Model includes baseline waist circumference, baseline HbA1c as covariates, baseline eGFR, geographic region, and treatment as fixed effects; Adjusted mean difference = -2.1, 95% CI 2-sided [-3.1 to -1.0], Standard Error of Mean 0.5
Statistical Analysis 2: Comparison: BI 10773 High (Drug Naive) vs Placebo (Drug Naive); Test type: Superiority or Other; p = 0.0015, ANCOVA — [p-value comment as in outcome 10, analysis 1]; Adjusted mean difference = -1.7, 95% CI 2-sided [-2.8 to -0.7], Standard Error of Mean 0.5
Statistical Analysis 3: Comparison: Placebo (Drug Naive) vs Sitagliptin 100mg (Drug Naive); Test type: Superiority or Other; p = 0.5052, ANCOVA — [p-value comment as in outcome 10, analysis 1]; Adjusted mean difference = 0.4, 95% CI 2-sided [-0.7 to 1.4], Standard Error of Mean 0.5
Statistical Analysis 4: Comparison: BI 10773 Low (Drug Naive) vs Sitagliptin 100mg (Drug Naive); Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 10, analysis 1]; Adjusted mean difference = -2.4, 95% CI 2-sided [-3.5 to -1.4], Standard Error of Mean 0.5
Statistical Analysis 5: Comparison: BI 10773 High (Drug Naive) vs Sitagliptin 100mg (Drug Naive); Test type: Superiority or Other; p = 0.0001, ANCOVA — [p-value comment as in outcome 10, analysis 1]; Adjusted mean difference = -2.1, 95% CI 2-sided [-3.1 to -1.0], Standard Error of Mean 0.5
Statistical Analysis 6: Comparison: BI 10773 Low (Pioglitazone) vs Placebo (Pioglitazone); Test type: Superiority or Other; p = 0.0064, ANCOVA — [p-value comment as in outcome 10, analysis 1]; Adjusted mean difference = -1.5, 95% CI 2-sided [-2.6 to -0.4], Standard Error of Mean 0.5
Statistical Analysis 7: Comparison: BI 10773 High (Pioglitazone) vs Placebo (Pioglitazone); Test type: Superiority or Other; p = 0.0642, ANCOVA — [p-value comment as in outcome 10, analysis 1]; Adjusted mean difference = -1.0, 95% CI 2-sided [-2.1 to 0.1], Standard Error of Mean 0.5
Statistical Analysis 8: Comparison: BI 10773 Low (Metformin) vs Placebo (Metformin); Test type: Superiority or Other; p = 0.0053, ANCOVA — [p-value comment as in outcome 10, analysis 1]; Adjusted mean difference = -1.0, 95% CI 2-sided [-1.8 to -0.3], Standard Error of Mean 0.4
Statistical Analysis 9: Comparison: BI 10773 High (Metformin) vs Placebo (Metformin); Test type: Superiority or Other; p < 0.0001, ANCOVA; Adjusted mean difference = -1.6, 95% CI 2-sided [-2.3 to -0.9], Standard Error of Mean 0.4
Statistical Analysis 10: Comparison: BI 10773 Low (Metformin+Sulfonylurea) vs Placebo (Metformin+Sulfonylurea); Test type: Superiority or Other; p = 0.0010, ANCOVA — [p-value comment as in outcome 10, analysis 1]; Adjusted mean difference = -1.3, 95% CI 2-sided [-2.1 to -0.6], Standard Error of Mean 0.4
Statistical Analysis 11: Comparison: BI 10773 High (Metformin+Sulfonylurea) vs Placebo (Metformin+Sulfonylurea); Test type: Superiority or Other; p = 0.0015, ANCOVA — [p-value comment as in outcome 10, analysis 1]; Adjusted mean difference = -1.3, 95% CI 2-sided [-2.1 to -0.5], Standard Error of Mean 0.4

11. Secondary Outcome: Waist Circumference (cm) Change From Baseline After 76 Weeks of Treatment
Description: Waist circumference (cm) - change from baseline after 76 weeks of treatment
Time Frame: Baseline and 76 weeks
Population: as for outcome 10
Measure: Least Squares Mean (Standard Error); unit: cm
Arm/Group | BI 10773 Low (Drug Naive) | BI 10773 High (Drug Naive) | Placebo (Drug Naive) | Sitagliptin 100mg (Drug Naive) | BI 10773 Low (Pioglitazone) | BI 10773 High (Pioglitazone) | Placebo (Pioglitazone) | BI 10773 Low (Metformin) | BI 10773 High (Metformin) | Placebo (Metformin) | BI 10773 Low (Metformin+Sulfonylurea) | BI 10773 High (Metformin+Sulfonylurea) | Placebo (Metformin+Sulfonylurea)
Number analyzed (Participants) | 223 | 224 | 228 | 221 | 163 | 167 | 165 | 216 | 213 | 207 | 222 | 215 | 219
cm | -1.5 (0.4) | -1.6 (0.4) | 0.1 (0.4) | 0.5 (0.4) | -1.4 (0.4) | -0.9 (0.4) | 0.0 (0.4) | -1.8 (0.3) | -1.3 (0.3) | -0.2 (0.3) | -1.6 (0.3) | -1.4 (0.3) | -0.3 (0.3)
Statistical Analysis 1: Comparison: BI 10773 Low (Drug Naive) vs Placebo (Drug Naive); Test type: Superiority or Other; p = 0.0028, ANCOVA — [p-value comment as in outcome 10, analysis 1]; Adjusted mean difference = -1.6, 95% CI 2-sided [-2.7 to -0.6], Standard Error of Mean 0.5
Statistical Analysis 2: Comparison: BI 10773 High (Drug Naive) vs Placebo (Drug Naive); Test type: Superiority or Other; p = 0.0019, ANCOVA — [p-value comment as in outcome 10, analysis 1]; Adjusted mean difference = -1.7, 95% CI 2-sided [-2.8 to -0.6], Standard Error of Mean 0.5
Statistical Analysis 3: Comparison: Placebo (Drug Naive) vs Sitagliptin 100mg (Drug Naive); Test type: Superiority or Other; p = 0.5044, ANCOVA — [p-value comment as in outcome 10, analysis 1]; Adjusted mean difference = 0.4, 95% CI 2-sided [-0.7 to 1.5], Standard Error of Mean 0.6
Statistical Analysis 4: Comparison: BI 10773 Low (Drug Naive) vs Sitagliptin 100mg (Drug Naive); Test type: Superiority or Other; p = 0.0003, ANCOVA — [p-value comment as in outcome 10, analysis 1]; Adjusted mean difference = -2.0, 95% CI 2-sided [-3.1 to -0.9], Standard Error of Mean 0.6
Statistical Analysis 5: Comparison: BI 10773 High (Drug Naive) vs Sitagliptin 100mg (Drug Naive); Test type: Superiority or Other; p = 0.0002, ANCOVA — [p-value comment as in outcome 10, analysis 1]; Adjusted mean difference = -2.1, 95% CI 2-sided [-3.2 to -1.0], Standard Error of Mean 0.6
Statistical Analysis 6: Comparison: BI 10773 Low (Pioglitazone) vs Placebo (Pioglitazone); Test type: Superiority or Other; p = 0.0109, ANCOVA — [p-value comment as in outcome 10, analysis 1]; Adjusted mean difference = -1.4, 95% CI 2-sided [-2.5 to -0.3], Standard Error of Mean 0.6
Statistical Analysis 7: Comparison: BI 10773 High (Pioglitazone) vs Placebo (Pioglitazone); Test type: Superiority or Other; p = 0.1238, ANCOVA — [p-value comment as in outcome 10, analysis 1]; Adjusted mean difference = -0.9, 95% CI 2-sided [-1.9 to 0.2], Standard Error of Mean 0.6
Statistical Analysis 8: Comparison: BI 10773 Low (Metformin) vs Placebo (Metformin); Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 10, analysis 1]; Adjusted mean difference = -1.6, 95% CI 2-sided [-2.4 to -0.8], Standard Error of Mean 0.4
Statistical Analysis 9: Comparison: BI 10773 High (Metformin) vs Placebo (Metformin); Test type: Superiority or Other; p = 0.0076, ANCOVA — [p-value comment as in outcome 10, analysis 1]; Adjusted mean difference = -1.1, 95% CI 2-sided [-1.9 to -0.3], Standard Error of Mean 0.4
Statistical Analysis 10: Comparison: BI 10773 Low (Metformin+Sulfonylurea) vs Placebo (Metformin+Sulfonylurea); Test type: Superiority or Other; p = 0.0049, ANCOVA — [p-value comment as in outcome 10, analysis 1]; Adjusted mean difference = -1.2, 95% CI 2-sided [-2.1 to -0.4], Standard Error of Mean 0.4
Statistical Analysis 11: Comparison: BI 10773 High (Metformin+Sulfonylurea) vs Placebo (Metformin+Sulfonylurea); Test type: Superiority or Other; p = 0.0178, ANCOVA — [p-value comment as in outcome 10, analysis 1]; Adjusted mean difference = -1.0, 95% CI 2-sided [-1.9 to -0.2], Standard Error of Mean 0.4

12. Secondary Outcome: Fasting Plasma Glucose Change From Baseline After 52 Weeks of Treatment
Description: Fasting plasma glucose - change from baseline after 52 weeks of treatment
Time Frame: Baseline and 52 weeks
Population: Full Analysis Set (FAS) which contained all randomised patients who received at least 1 dose of study drug and had a baseline fasting plasma glucose assessment, irrespective of participation in the extension trial -LOCF
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | BI 10773 Low (Drug Naive) | BI 10773 High (Drug Naive) | Placebo (Drug Naive) | Sitagliptin 100mg (Drug Naive) | BI 10773 Low (Pioglitazone) | BI 10773 High (Pioglitazone) | Placebo (Pioglitazone) | BI 10773 Low (Metformin) | BI 10773 High (Metformin) | Placebo (Metformin) | BI 10773 Low (Metformin+Sulfonylurea) | BI 10773 High (Metformin+Sulfonylurea) | Placebo (Metformin+Sulfonylurea)
Number analyzed (Participants) | 223 | 223 | 226 | 223 | 163 | 168 | 165 | 216 | 213 | 207 | 225 | 215 | 224
mg/dL | -18.9 (2.0) | -23.9 (2.0) | 13.3 (2.0) | -3.9 (2.0) | -16.7 (2.8) | -20.7 (2.8) | 10.3 (2.8) | -16.7 (1.9) | -19.7 (1.9) | 7.6 (2.0) | -18.4 (2.1) | -19.3 (2.1) | 9.4 (2.1)
Statistical Analysis 1: Comparison: BI 10773 Low (Drug Naive) vs Placebo (Drug Naive); Test type: Superiority or Other; p < 0.0001, ANCOVA — Model includes baseline fasting plasma glucose, baseline HbA1c as covariates, baseline eGFR, geographic region, and treatment as fixed effects; Adjusted mean difference = -32.3, 95% CI 2-sided [-37.8 to -26.7], Standard Error of Mean 2.8
Statistical Analysis 2: Comparison: BI 10773 High (Drug Naive) vs Placebo (Drug Naive); Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 12, analysis 1]; Adjusted mean difference = -37.2, 95% CI 2-sided [-42.8 to -31.7], Standard Error of Mean 2.8
Statistical Analysis 3: Comparison: Placebo (Drug Naive) vs Sitagliptin 100mg (Drug Naive); Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 12, analysis 1]; Adjusted mean difference = -17.3, 95% CI 2-sided [-22.9 to -11.7], Standard Error of Mean 2.8
Statistical Analysis 4: Comparison: BI 10773 Low (Drug Naive) vs Sitagliptin 100mg (Drug Naive); Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 12, analysis 1]; Adjusted mean difference = -15.0, 95% CI 2-sided [-20.6 to -9.4], Standard Error of Mean 2.9
Statistical Analysis 5: Comparison: BI 10773 High (Drug Naive) vs Sitagliptin 100mg (Drug Naive); Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 12, analysis 1]; Adjusted mean difference = -19.9, 95% CI 2-sided [-25.5 to -14.4], Standard Error of Mean 2.8
Statistical Analysis 6: Comparison: BI 10773 Low (Pioglitazone) vs Placebo (Pioglitazone); Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 12, analysis 1]; Adjusted mean difference = -27.1, 95% CI 2-sided [-35.0 to -19.2], Standard Error of Mean 4.0
Statistical Analysis 7: Comparison: BI 10773 High (Pioglitazone) vs Placebo (Pioglitazone); Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 12, analysis 1]; Adjusted mean difference = -31.0, 95% CI 2-sided [-38.9 to -23.2], Standard Error of Mean 4.0
Statistical Analysis 8: Comparison: BI 10773 Low (Metformin) vs Placebo (Metformin); Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 12, analysis 1]; Adjusted mean difference = -24.3, 95% CI 2-sided [-29.7 to -18.9], Standard Error of Mean 2.7
Statistical Analysis 9: Comparison: BI 10773 High (Metformin) vs Placebo (Metformin); Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 12, analysis 1]; Adjusted mean difference = -27.3, 95% CI 2-sided [-32.7 to -21.9], Standard Error of Mean 2.8
Statistical Analysis 10: Comparison: BI 10773 Low (Metformin+Sulfonylurea) vs Placebo (Metformin+Sulfonylurea); Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 12, analysis 1]; Adjusted mean difference = -27.8, 95% CI 2-sided [-33.6 to -22.0], Standard Error of Mean 2.9
Statistical Analysis 11: Comparison: BI 10773 High (Metformin+Sulfonylurea) vs Placebo (Metformin+Sulfonylurea); Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 12, analysis 1]; Adjusted mean difference = -28.7, 95% CI 2-sided [-34.5 to -22.8], Standard Error of Mean 3.0

13. Secondary Outcome: Fasting Plasma Glucose Change From Baseline After 76 Weeks of Treatment
Description: Fasting plasma glucose - change from baseline after 76 weeks of treatment
Time Frame: Baseline and 76 weeks
Population: as for outcome 12
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | BI 10773 Low (Drug Naive) | BI 10773 High (Drug Naive) | Placebo (Drug Naive) | Sitagliptin 100mg (Drug Naive) | BI 10773 Low (Pioglitazone) | BI 10773 High (Pioglitazone) | Placebo (Pioglitazone) | BI 10773 Low (Metformin) | BI 10773 High (Metformin) | Placebo (Metformin) | BI 10773 Low (Metformin+Sulfonylurea) | BI 10773 High (Metformin+Sulfonylurea) | Placebo (Metformin+Sulfonylurea)
Number analyzed (Participants) | 223 | 223 | 226 | 223 | 163 | 168 | 165 | 216 | 213 | 207 | 225 | 215 | 224
mg/dL | -17.2 (2.1) | -20.4 (2.1) | 14.4 (2.1) | -1.8 (2.1) | -13.9 (2.9) | -18.0 (2.9) | 9.4 (2.9) | -14.5 (2.0) | -20.9 (2.0) | 10.5 (2.0) | -19.5 (2.2) | -20.4 (2.2) | 11.4 (2.2)
Statistical Analysis 1: Comparison: BI 10773 Low (Drug Naive) vs Placebo (Drug Naive); Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 12, analysis 1]; Adjusted mean difference = -31.7, 95% CI 2-sided [-37.4 to -25.9], Standard Error of Mean 2.9
Statistical Analysis 2: Comparison: BI 10773 High (Drug Naive) vs Placebo (Drug Naive); Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 12, analysis 1]; Adjusted mean difference = -34.9, 95% CI 2-sided [-40.7 to -29.1], Standard Error of Mean 2.9
Statistical Analysis 3: Comparison: Placebo (Drug Naive) vs Sitagliptin 100mg (Drug Naive); Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 12, analysis 1]; Adjusted mean difference = -16.3, 95% CI 2-sided [-22.1 to -10.5], Standard Error of Mean 3.0
Statistical Analysis 4: Comparison: BI 10773 Low (Drug Naive) vs Sitagliptin 100mg (Drug Naive); Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 12, analysis 1]; Adjusted mean difference = -15.4, 95% CI 2-sided [-21.2 to -9.6], Standard Error of Mean 3.0
Statistical Analysis 5: Comparison: BI 10773 High (Drug Naive) vs Sitagliptin 100mg (Drug Naive); Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 12, analysis 1]; Adjusted mean difference = -18.7, 95% CI 2-sided [-24.5 to -12.8], Standard Error of Mean 3.0
Statistical Analysis 6: Comparison: BI 10773 Low (Pioglitazone) vs Placebo (Pioglitazone); Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 12, analysis 1]; Adjusted mean difference = -23.3, 95% CI 2-sided [-31.4 to -15.3], Standard Error of Mean 4.1
Statistical Analysis 7: Comparison: BI 10773 High (Pioglitazone) vs Placebo (Pioglitazone); Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 12, analysis 1]; Adjusted mean difference = -27.4, 95% CI 2-sided [-35.4 to -19.4], Standard Error of Mean 4.1
Statistical Analysis 8: Comparison: BI 10773 Low (Metformin) vs Placebo (Metformin); Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 12, analysis 1]; Adjusted mean difference = -25.1, 95% CI 2-sided [-30.5 to -19.6], Standard Error of Mean 2.8
Statistical Analysis 9: Comparison: BI 10773 High (Metformin) vs Placebo (Metformin); Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 12, analysis 1]; Adjusted mean difference = -31.4, 95% CI 2-sided [-36.9 to -25.9], Standard Error of Mean 2.8
Statistical Analysis 10: Comparison: BI 10773 Low (Metformin+Sulfonylurea) vs Placebo (Metformin+Sulfonylurea); Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 12, analysis 1]; Adjusted mean difference = -31.0, 95% CI 2-sided [-37.0 to -24.9], Standard Error of Mean 3.1
Statistical Analysis 11: Comparison: BI 10773 High (Metformin+Sulfonylurea) vs Placebo (Metformin+Sulfonylurea); Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 12, analysis 1]; Adjusted mean difference = -31.8, 95% CI 2-sided [-37.9 to -25.7], Standard Error of Mean 3.1

ADVERSE EVENTS:
Time Frame: From signing of the informed consent until 7 days (inclusive) after last treatment
Description: For all safety analyses (except drug-related AEs), patients are assigned to the treatment group "as treated" at inclusion (if a patient erroneously receives the wrong trial drug, the patient is analysed as per the first treatment received). For drug-related AEs, patients are assigned to the actual treatment at onset of AE.
Groups:
- Placebo (Metformin+Sulfonylurea): Patients rolled over from 1245.23
  Placebo tablets matching Empagliflozin
  Placebo: Placebo matching Empagliflozin 10 mg
  Placebo: Placebo matching Empagliflozin 25 mg
Arm/Group | Empagliflozin 10 mg (Drug Naive) | Empagliflozin 25 mg (Drug Naive) | Placebo (Drug Naive) | Sitagliptin 100mg (Drug Naive) | Empagliflozin 10 mg (Pioglitazone) | Empagliflozin 25 mg (Pioglitazone) | Placebo (Pioglitazone) | Empagliflozin 10 mg (Metformin) | Empagliflozin 25 mg (Metformin) | Placebo (Metformin) | Empagliflozin 10 mg (Metformin+Sulfonylurea) | Empagliflozin 25 mg (Metformin+Sulfonylurea) | Placebo (Metformin+Sulfonylurea)
Serious Adverse Events (participants affected / at risk) | 23/229 | 25/224 | 16/223 | 18/223 | 11/165 | 13/165 | 15/168 | 24/206 | 19/217 | 17/214 | 31/225 | 29/224 | 24/217
Other Adverse Events (participants affected / at risk) | 134/229 | 110/224 | 92/223 | 116/223 | 110/165 | 96/165 | 107/168 | 122/206 | 113/217 | 106/214 | 146/225 | 147/224 | 142/217
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Empagliflozin 10 mg (Drug Naive) (N=229) | Empagliflozin 25 mg (Drug Naive) (N=224) | Placebo (Drug Naive) (N=223) | Sitagliptin 100mg (Drug Naive) (N=223) | Empagliflozin 10 mg (Pioglitazone) (N=165) | Empagliflozin 25 mg (Pioglitazone) (N=165) | Placebo (Pioglitazone) (N=168) | Empagliflozin 10 mg (Metformin) (N=206) | Empagliflozin 25 mg (Metformin) (N=217) | Placebo (Metformin) (N=214) | Empagliflozin 10 mg (Metformin+Sulfonylurea) (N=225) | Empagliflozin 25 mg (Metformin+Sulfonylurea) (N=224) | Placebo (Metformin+Sulfonylurea) (N=217)
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Amoebic colitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cervicitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dengue fever (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pseudomonas infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pyelonephritis acute (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Septic shock (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Urosepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Anal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gangrene (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Atypical pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cytomegalovirus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Genital infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Herpes virus infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infected skin ulcer (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Listeria sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Peritonitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary tuberculosis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Salmonellosis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Schistosomiasis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ovarian neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rectosigmoid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Anaplastic large cell lymphoma T- and null-cell types (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Breast cancer female (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastrooesophageal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Empty sella syndrome (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Goitre (Endocrine disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Hyperparathyroidism (Endocrine disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lactic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Insulin-requiring type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Stress (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cerebral infarction (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Brain stem infarction (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Carotid artery stenosis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Brain stem stroke (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Carotid artery disease (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cerebral ischaemia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Diabetic neuropathy (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Lacunar infarction (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Radiculitis brachial (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Trigeminal neuralgia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Carpal tunnel syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cervicobrachial syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Convulsion (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Intercostal neuralgia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vascular headache (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vertebrobasilar insufficiency (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diabetic retinopathy (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cataract (Eye disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dacryostenosis acquired (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Glaucoma (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lens dislocation (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Retinal detachment (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Retinal vein occlusion (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vitreous haemorrhage (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vertigo positional (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sudden hearing loss (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Meniere's disease (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Coronary artery disease (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 2 | 2 | 1 | 0 | 1 | 1
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 2 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 1
Arteriosclerosis coronary artery (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Angina unstable (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Atrial flutter (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cardio-respiratory arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Congestive cardiomyopathy (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0
Prinzmetal angina (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Aortic valve stenosis (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Stress cardiomyopathy (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ventricular tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardiogenic shock (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Left ventricular failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute left ventricular failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0
Femoral artery occlusion (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vascular calcification (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vascular occlusion (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ischaemia (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Arterial occlusive disease (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Venous occlusion (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Upper airway resistance syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Haemorrhoids (Gastrointestinal disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anal fissure (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oesophageal rupture (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastric polyps (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Colitis ulcerative (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Duodenal ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Faecaloma (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Large intestine polyp (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Liver injury (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatitis toxic (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cirrhosis alcoholic (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Liver disorder (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Jaundice (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 1 | 1 | 1 | 0 | 2
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Osteoarthropathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Femoroacetabular impingement (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Plica syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Synovitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tenosynovitis stenosans (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Facet joint syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 2 | 1 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Diabetic nephropathy (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Renal tubular necrosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cystitis haemorrhagic (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypotonic urinary bladder (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Polyuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Endometrial hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Breast mass (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Menorrhagia (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gilbert's syndrome (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hydrocele (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Phimosis (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Syringomyelia (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1
Death (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chest discomfort (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hernia (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Impaired healing (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sudden death (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemoglobin decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Smear cervix abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Comminuted fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 0
Hand fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injury (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Traumatic fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ligament rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Animal bite (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Multiple fractures (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Neck injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Post-traumatic neck syndrome (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Knee arthroplasty (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hip arthroplasty (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Photocoagulation (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vitrectomy (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Leg amputation (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Empagliflozin 10 mg (Drug Naive) (N=229) | Empagliflozin 25 mg (Drug Naive) (N=224) | Placebo (Drug Naive) (N=223) | Sitagliptin 100mg (Drug Naive) (N=223) | Empagliflozin 10 mg (Pioglitazone) (N=165) | Empagliflozin 25 mg (Pioglitazone) (N=165) | Placebo (Pioglitazone) (N=168) | Empagliflozin 10 mg (Metformin) (N=206) | Empagliflozin 25 mg (Metformin) (N=217) | Placebo (Metformin) (N=214) | Empagliflozin 10 mg (Metformin+Sulfonylurea) (N=225) | Empagliflozin 25 mg (Metformin+Sulfonylurea) (N=224) | Placebo (Metformin+Sulfonylurea) (N=217)
Urinary tract infection (Infections and infestations) | 21 | 20 | 13 | 18 | 33 | 29 | 33 | 23 | 25 | 18 | 28 | 33 | 33
Nasopharyngitis (Infections and infestations) | 27 | 32 | 25 | 27 | 7 | 10 | 9 | 39 | 36 | 29 | 24 | 36 | 34
Upper respiratory tract infection (Infections and infestations) | 12 | 17 | 16 | 19 | 11 | 9 | 15 | 17 | 7 | 21 | 24 | 18 | 21
Bronchitis (Infections and infestations) | 10 | 11 | 6 | 12 | 2 | 5 | 4 | 8 | 6 | 6 | 8 | 12 | 8
Influenza (Infections and infestations) | 9 | 6 | 6 | 6 | 4 | 0 | 4 | 5 | 4 | 6 | 4 | 7 | 11
Anaemia (Blood and lymphatic system disorders) | 8 | 2 | 2 | 0 | 13 | 7 | 11 | 5 | 2 | 3 | 5 | 1 | 4
Hyperglycaemia (Metabolism and nutrition disorders) | 63 | 20 | 11 | 28 | 49 | 27 | 23 | 56 | 25 | 14 | 59 | 24 | 26
Hypoglycaemia (Metabolism and nutrition disorders) | 3 | 4 | 2 | 2 | 8 | 4 | 7 | 8 | 15 | 10 | 40 | 53 | 46
Dyslipidaemia (Metabolism and nutrition disorders) | 15 | 16 | 14 | 14 | 26 | 23 | 21 | 7 | 16 | 8 | 5 | 5 | 5
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 6 | 3 | 9 | 7 | 1 | 2 | 2 | 1 | 0 | 2
Dizziness (Nervous system disorders) | 6 | 6 | 6 | 7 | 6 | 6 | 14 | 6 | 5 | 4 | 16 | 13 | 17
Headache (Nervous system disorders) | 9 | 10 | 6 | 5 | 8 | 10 | 13 | 7 | 6 | 7 | 13 | 17 | 10
Hypertension (Vascular disorders) | 12 | 11 | 5 | 14 | 16 | 6 | 3 | 6 | 7 | 11 | 2 | 6 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 9 | 3 | 6 | 6 | 4 | 3 | 7 | 5 | 7 | 3 | 13 | 6
Dyspepsia (Gastrointestinal disorders) | 2 | 1 | 2 | 2 | 2 | 10 | 4 | 2 | 3 | 2 | 4 | 3 | 4
Diarrhoea (Gastrointestinal disorders) | 9 | 12 | 6 | 8 | 5 | 6 | 4 | 10 | 10 | 9 | 7 | 10 | 7
Back pain (Musculoskeletal and connective tissue disorders) | 11 | 7 | 7 | 18 | 9 | 9 | 7 | 10 | 9 | 11 | 11 | 15 | 12
Arthralgia (Musculoskeletal and connective tissue disorders) | 11 | 9 | 10 | 7 | 9 | 10 | 10 | 5 | 7 | 7 | 4 | 11 | 8
Glycosylated haemoglobin increased (Investigations) | 9 | 10 | 1 | 6 | 8 | 3 | 2 | 9 | 6 | 2 | 12 | 6 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.